# Official Title of Study:

An Investigational Study to Evaluate Experimental Medication BMS-986165 Compared to Placebo in Participants With Plaque Psoriasis (POETYK-PSO-3) in Mainland China, Taiwan, and South Korea (POETYK-PSO-3)

NCT Number: NCT04167462

Document Date (Date in which document was last revised): 11-Nov-2020

Page: 1

Protocol Number: IM011065
IND Number: 131,993
EX-US Non-IND
EUDRACT Number: N/A

Date: 11-Nov-2020

Revised Protocol 05, Final Approved

# **Clinical Protocol IM011065:**

A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Subjects With Moderate-to-Severe Plaque Psoriasis

Short Title: Efficacy and Safety of BMS-986165 versus Placebo in Subjects with Plaque Psoriasis

### **Revised Protocol 05**

Site Number: All sites in Mainland China, Taiwan, and South Korea



### 24-hr Emergency Telephone Number

North America:

Asia Pacific:

### **Bristol-Myers Squibb Research and Development**

3401 Princeton Pike Lawrenceville, NJ 08648 Avenue de Finlande 4 B-1420 Braine-l'Alleud, Belgium 6-5-1 Nishi-Shinjuku, Shinjuku-ku, Tokyo, 163-1328, Japan

This document is the confidential and proprietary information of Bristol-Myers Squibb Company and its global affiliates (BMS). By reviewing this document, you agree to keep it confidential and to use and disclose it solely for the purpose of assessing whether your organization will participate in and/or the performance of the proposed BMS sponsored study. Any permitted disclosures will be made only on a confidential "need to know" basis

within your organization or to your independent ethics committee(s). Any other use, copying, disclosure or dissemination of this information is strictly prohibited unless expressly authorized in writing by BMS. Any supplemental information (eg, amendments) that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this document. Any person who receives this document without due authorization from BMS is requested to return it to BMS or promptly destroy it. All other rights reserved. References to BMS in this protocol may apply to partners to which BMS has transferred obligations, eg, a Contract Research Organization (CRO).

# **DOCUMENT HISTORY**

| Document | Date of Issue | Approver(s) | Summary of Change |
|---|---|---|---|
| Revised<br>Protocol 05<br>(im011065-<br>revprot05) | 11-Nov-2020 | | -Added a Week 16 database lock so the analysis of the efficacy and safety data collected up to Week 16 could be performed after the double-blind portion of the study is complete |
| | | | -Clarified the unblinding procedures for personnel performing the Week 16 primary endpoint analysis |
| Revised Protocol 03b South Korea— specific (Revised Protocol 05 <sup>a</sup> ) | 18-Sept-2020 | | Korea-Specific Revised<br>Protocol - Included changes<br>listed above for the Global<br>Revised Protocol 04 |
| (im011065-<br>revprot03b-sk-<br>specific) | | | |
| Revised<br>Protocol 04 | 19-Jun-2020 | | -Provided clarifications in<br>the protocol to aid sites and<br>subjects in the conduct of<br>the study |
| (im011065-<br>revprot04) | | | -Updated sample size from 180 subjects to approximately 219 subjects |
| | | | -Added and updated<br>relevant protocol deviation<br>criteria for the Per Protocol<br>Set |
| | | | -Corrected typographical errors |
| | | | -In the set of subgroup<br>analyses for the coprimary<br>efficacy endpoints, added a<br>new analysis for systemic<br>treatment-naïve subjects. |

| Document | Date of Issue | Approver(s) | Summary of Change |
|---|---|---|---|
| Revised Protocol 03a South Korea— specific (Revised Protocol 04 <sup>a</sup> ) (im011065- revprot03a-sk- specific) | 05-Jul-2019 | | South Korea–specific<br>Revised Protocol to include<br>HBV DNA monitoring<br>plans for subjects who are<br>HBsAg-, and HBsAb+<br>and/or HBcAb+. |
| Revised Protocol 03 (Amendment 03 <sup>a</sup> ) (im011065- revprot03) | 24 June 2019 | | -Updated the Sponsor's contact information, made typographic corrections to the protocol, and revised certain exclusion criteria to be consistent with certain elements of the Phase 2 study of BMS-986165 in psoriasis as well as other Phase 3 studies in psoriasisUpdated text in the definition of sPGA in Section 8.1.1.1 to be consistent with the description in Appendix 5. -Removed 'change from baseline in DLQI score.' The reason for this change is that DLQI endpoint 'DLQI 0/1 among subjects with baseline DLQI score ≥2' is clinically meaningful and is already in the hierarchy. |

| Document | Date of Issue | Approver(s) | Summary of Change |
|---|---|---|---|
| Revised Protocol 02 (Amendment 02a) (im011065- revprot02) | 09 April 2019 | | Includes modifications to protocol sections affected by removal of sites in Singapore, where the -065 study will no longer be conducted. Overall, the subject population will remain at 180 subjects and enrollment will be competitive. |
| Revised Protocol 01 (Amendment 01a) (im011065- revprot01) | 03 December<br>2018 | | Includes modifications to protocol sections affected by the addition to this mainland China-specific study of one region (Taiwan) and two countries where the -065 study will also be conducted (Singapore and South Korea). Overall, the subject population will remain at 180 subjects and enrollment will be competitive. |
| Original<br>Protocol<br>(im011065-<br>prot) | 22 June 2018 | | N/A |

<sup>&</sup>lt;sup>a</sup> Document naming conventions have been updated. Legacy numbering is provided for consistency.

Clinical Protocol BMS-986165

# **OVERALL RATIONALE FOR REVISED PROTOCOL 05:** Rationale:

The primary purpose of this global revised protocol is to provide clarifications in the protocol to aid sites and subjects in the conduct of the study.

Key modifications and clarifications are summarized as follows:

- Added a Week 16 database lock so the analysis of the efficacy and safety data collected up to Week 16 could be performed after the double-blind portion of the study is complete
- Clarified the unblinding procedures for personnel performing the Week 16 primary endpoint analysis

Substantive changes made to the previous version of the global protocol and the rationale for these changes are noted below in the summary of key changes table. All changes applied to the protocol body were applied to the synopsis, as necessary; synopsis changes are not included in the summary of key changes table. Only major additions and deletions are provided in this summary document; all minor grammatical, formatting, stylistic changes, or clarifications as well as organizational changes are not included.

| SUMMARY O | F KEY CHANGES FOR REVISED PROTOCOL | 05: |
|---|---|---|
| <b>Protocol Section</b> | Revised Protocol Text | Rationale for Change |
| Study<br>Acknowledgment<br>/Disclosure | This page was removed. | To conform to the BMS protocol model document, this page is now provided as a standalone document. |
| 1 2 Cabadala af | Updated row in Table 1 (Screening Procedures): Fasting Lipid Panel | Clarified that the lipid panel in the Screening Procedures |
| 1.3 Schedule of Activities | Added text in the Notes column for this row: Subjects are required to fast for at least 10 hours prior to collection. | should be performed after the<br>subject has fasted for<br>10 hours, like other lipid<br>panels in the study |
| 9.4 Efficacy<br>Analyses<br>9.4.1.2<br>Sensitivity<br>Analyses for the<br>Coprimary<br>Endpoints<br>9.6.3 Relevant<br>Protocol<br>Deviations | Updated text in Section 9.4: Details of the planned analyses of endpoints during the 16-week double-blind placebo-controlled period will be documented in the statistical analysis plan (SAP) and finalized before <b>the Week 16</b> database lock. Updated text in Section 9.4.1.2: | Clarified that the database lock mentioned in each section refers to the newly added Week 16 database lock |

| SUMMARY OF KEY CHANGES FOR REVISED PROTOCOL05: | | |
|---|---|---|
| <b>Protocol Section</b> | Revised Protocol Text | Rationale for Change |
| | Sensitivity analyses to be performed for the coprimary endpoints will be described in the SAP prior to <b>the Week 16</b> database lock. | |
| | Updated text in Section 9.6.3: | |
| | All subjects with relevant protocol deviations will be identified prior to <b>the Week 16</b> database lock. | |
| 6.3.3 Unblinding<br>for Week 16<br>Primary Endpoint<br>Analysis | An unblinded analysis of data through Week 16 will be performed after all subjects complete their Week 16 visit or have discontinued prior to Week 16. A select group of personnel who are not involved in the conduct of the study will review the results to write a clinical study report. Following the Week 16 analysis until the end of the study, the investigators, subjects, and clinical trial team members who directly cooperate with the site staff will continue to remain blinded to the initial treatment assignment. Details of maintaining the blind following the unblinded analysis will be finalized prior to the Week 16 database lock. A final analysis will be performed after all subjects complete the Week 52 visit or discontinue prior to the Week 52 visit, and a clinical study report will be written. | Clarified the unblinding procedures for the personnel performing the Week 16 primary endpoint analysis |
| 9.8 Analysis and<br>Reporting | Added section: An unblinded analysis of the data collected up to Week 16 will be conducted once all randomized subjects have either completed the placebo-controlled treatment period (ie, through Week 16) or have discontinued prior to Week 16. Details of these analyses will be provided in an SAP that will be finalized before the Week 16 database lock. A final database lock and analysis will occur after all subjects complete Week 52 or discontinue prior to Week 52. | Added a Week 16 database lock so the analysis of the efficacy and safety data collected up to Week 16 could be performed after the double-blind portion of the study is complete |

# TABLE OF CONTENTS

| TITLE PAGE | 1 |
|--------------------------------------------------------------|-----|
| TABLE OF CONTENTS | 8 |
| 11 APPENDICES | 75 |
| APPENDIX 1 ABBREVIATIONS AND TRADEMARKS | 76 |
| APPENDIX 2 STUDY GOVERNANCE CONSIDERATIONS | 80 |
| APPENDIX 3 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS | |
| DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, | |
| FOLLOW-UP, AND REPORTING | 88 |
| APPENDIX 4 WOMEN OF CHILDBEARING POTENTIAL DEFINTIONS AND | |
| METHODS OF CONTRACEPTION | 92 |
| APPENDIX 5 STATIC PHYSICIAN'S GLOBAL ASSESSMENT OF PSORIASIS | |
| (SPGA) | 96 |
| APPENDIX 6 PSORIASIS AREA AND SEVERITY INDEX (PASI) | 97 |
| APPENDIX 7 SCALP-SPECIFIC PHYSICIAN'S GLOBAL ASSESSMENT | |
| (SSPGA) | 98 |
| APPENDIX 9 PHYSICIAN'S GLOBAL ASSESSMENT-FINGERNAILS (PGA-F) | |
| | 100 |
| APPENDIX 11 PALMOPLANTAR PSORIASIS PHYSICIAN'S GLOBAL | |
| ASSESSMENT (PP-PGA) | 103 |
| | 105 |
| APPENDIX 13 PSORIASIS SYMPTOMS AND SIGNS DIARY (PSSD) | 105 |
| APPENDIX 14 DERMATOLOGY LIFE QUALITY INDEX (DLQI) | 106 |
| APPENDIX 20 PSORIATIC ARTHRITIS SCREENING AND EVALUATION | 440 |
| (PASE) QUESTIONNAIRE | 119 |
| APPENDIX 21 EIGHT-ITEM PATIENT HEALTH QUESTIONNAIRE (PHQ-8) | 121 |
| APPENDIX 22 SUICIDAL IDEATION AND BEHAVIOR CATEGORIES AND | |
| DEFINITIONS | 122 |

#### 1 PROTOCOL SUMMARY

### 1.1 Synopsis

**Protocol Title:** A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Subjects with Moderate-to-Severe Plaque Psoriasis

Short Title: Efficacy and Safety of BMS-986165 versus Placebo in Subjects with Plaque Psoriasis

**Study Phase: 3** 

#### **Rationale:**

BMS-986165 is being evaluated as a therapeutic option for the treatment of subjects with moderate-to-severe plaque psoriasis based on results of a recently completed 12-week, randomized, Phase 2, placebo-controlled, parallel-group study (Study IM011011). The Phase 2 study was conducted with the following 5 different BMS-986165 treatment arms: 3 mg every other day (QOD); 3 mg once daily (QD); 3 mg twice daily (BID); 6 mg BID; and 12 mg QD. Overall, 267 subjects were randomized (44 to 45 subjects per treatment arm) in the Phase 2 study. All BMS-986165 treatment groups, except 3 mg QOD, achieved the primary endpoint of superiority compared to placebo in the proportion of subjects experiencing at least a 75% improvement in the Psoriasis Area and Severity Index (PASI 75) after 12 weeks of treatment. Compared with the placebo treatment group (6.7%), 38.6% (p = 0.0003), 68.9% (p < 0.0001), 66.7% (p < 0.0001) and 75% (p < 0.0001) of the subjects treated with BMS-986165 at 3 mg QD, 3 mg BID, 6 mg BID and 12 mg QD doses achieved a PASI 75 response respectively. The PASI 75 responses appear to plateau at the dose of 3 mg BID. The Phase 3 IM011065 study is designed to confirm the efficacy and safety of BMS-986165 6 mg QD, which is expected to have equivalent efficacy as the 3 mg BID dose in Phase 2, in a population of subjects with stable moderate-to-severe plaque psoriasis.

### **Study Population:**

Study IM011065 will enroll subjects in mainland China, Taiwan, and South Korea. Men and women  $\geq$ 18 years of age diagnosed with stable (defined as no morphology changes or significant flares of disease activity in the opinion of the investigator) plaque psoriasis for  $\geq$ 6 months and with moderate-to-severe disease characterized by involvement of  $\geq$ 10% of body surface area (BSA), static Physician's Global Assessment (sPGA)  $\geq$ 3, and a PASI score  $\geq$ 12, and who are candidates for phototherapy or systemic therapy (Section 5.1) will be eligible to participate in the study.

### **Objectives and Endpoints:**

| Objective | Endpoint |
|---|---|
| Primary | |
| <ul> <li>Assess whether BMS-986165 is superior to<br/>placebo at Week 16 in the treatment of subjects<br/>with moderate-to-severe plaque psoriasis</li> </ul> | <ul><li>sPGA 0/1</li><li>PASI 75</li></ul> |
| Selected Secondary Endpoints | |
| | • sPGA 0/1 |
| • Assess whether BMS-986165 is superior to placebo over the first 16 weeks of treatment | <ul> <li>PASI 90</li> <li>sPGA 0</li> <li>PASI 100</li> </ul> |
| Evaluate improvement in patient reported outcomes for BMS-986165 compared with placebo through Week 16 | <ul> <li>Change from baseline in Psoriasis Symptoms and Signs Diary (PSSD) symptom score</li> <li>PSSD symptom score of 0 (among subjects with a baseline PSSD symptom score ≥1)</li> </ul> |

### **Overall Design:**

This will be a 52 week, multicenter, randomized, double-blind, placebo-controlled study in subjects with stable moderate-to-severe plaque psoriasis. Subjects will undergo screening evaluations within 28 days prior to administration of study treatment to determine eligibility. Following the screening process, approximately 219 subjects will be randomized in a 2:1 ratio to either BMS-986165 6 mg QD or placebo, respectively.

Randomization should not occur until at least 8 days after the screening visit to allow collection of PSSD data during screening in order to calculate a baseline PSSD score. Randomization will be stratified by country (mainland China vs. non-mainland China) and previous biologic use (for psoriasis, psoriatic arthritis or other inflammatory diseases only; yes/no).

At Week 16, subjects randomized to placebo from screening through the Week 16 visit will be switched to BMS-986165 6 mg QD through Week 52 in a blinded manner, so that subjects who had been randomized to placebo will not know if they had been randomized to BMS-986165 or to

placebo post-screening. Subjects randomized to BMS-986165 6 mg QD will continue their current dose through Week 52.

At Week 24, a subject with sPGA  $\geq$ 3 may be treated with restricted topical medications, such as topical high potency corticosteroids (WHO Classes I-V) but only at this time point and at the discretion of the investigator. This treatment may be continued through end of study.

Subjects who discontinue study treatment early are expected to remain in the study for continued follow-up until Week 52.

Subjects completing 52 weeks of treatment may be eligible to roll over to a separate long-term extension study and be treated with open-label BMS-986165 6 mg QD.

Subjects who choose not to roll over to the long-term extension study at Week 52 will be followed up for safety for 4 additional weeks, from Week 52 through Week 56.

### **Treatment Arms and Duration:**

**Study treatment:** Subjects in both treatment groups will take oral doses of one of the investigational product (IP), either BMS-986165 or placebo QD, for 16 weeks. After Week 16, all subjects will receive BMS-986165.

| Study Drug for Study IM011065 | | |
|-------------------------------|------|----|
| Medication Potency IP/Non-IP | | |
| BMS-986165 tablet | 6 mg | IP |
| placebo tablet | n/a | IP |

<sup>•</sup> IP = Investigational Product; n/a = not applicable.

### **Statistical Methods:**

### General Methodology

The primary efficacy analysis population will be the Full Analysis Set (FAS). The FAS will include all subjects who were randomized to receive assigned study treatment.

The analysis model for the coprimary efficacy endpoints and secondary binary endpoints will use stratified Cochran-Mantel-Haenszel (CMH) tests stratified by country (mainland China vs. non-mainland China) and previous biologic treatment use for psoriasis, psoriatic arthritis or other inflammatory disease (yes/no) to compare the response rates of BMS-986165 6 mg QD to placebo (see also Section 4.1.2). Nonresponder imputation will be used for binary endpoints for subjects who discontinue early, start a protocol prohibited medication/therapy that could improve psoriasis, or who have otherwise missing endpoint data prior to the specified timepoint.

The analysis model for continuous secondary endpoints will use analysis of covariance (ANCOVA) with treatment and previous biologic treatment use for psoriasis, psoriatic arthritis or other inflammatory disease (yes/no) as fixed effects. The baseline value will be added to the model

as a covariate. Treatment differences based on least-squares (LS) means and the corresponding 2-sided 95% confidence intervals (CIs) will be provided for the difference between BMS-986165 6 mg QD and placebo for each endpoint being assessed.

# Testing Strategy for Efficacy Endpoints

The primary family of coprimary endpoints will each be tested at a probability of making a Type I error of 0.05 first, and if significant for both endpoints, testing will proceed for the secondary family of key secondary endpoints. The primary family of coprimary endpoints will be the serial gatekeeper for proceeding with testing of the secondary family of key secondary efficacy endpoints.

Primary Family – Coprimary endpoints compared with placebo; both must be significant at the probability of making a Type I error of 0.05 in order to proceed with the secondary family tests for the key secondary endpoints:

- Primary 1: Proportion of subjects who achieve sPGA 0/1 at Week 16
- Primary 2: Proportion of subjects who achieve PASI 75 at Week 16

In order to control for Type I error rate inflation within the secondary family of key secondary endpoints, a hierarchical testing method will be implemented for the key secondary endpoints. A hierarchical test may only proceed to the next key secondary endpoint if the null hypothesis is rejected at a probability of making a Type I error of 0.05. If an endpoint fails at any step, then all subsequent p-values will be considered descriptive.

### Safety Analysis

Safety data will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) for continuous variables and frequency distributions (counts and percentages) for categorical variables.

Clinical Protocol BMS-986165

### 1.2 Schema



QD = once daily

The coprimary endpoints will be evaluated at Week 16. The duration of the study for each participant will be up to 52 weeks on treatment and 4 additional weeks for safety follow-up.

# 1.3 Schedule of Activities (SOA)

The schedules of assessments and procedures are documented in Table 1 for screening, Table 2 for baseline through Week 20, and Table 3 for Week 24 through Week 52.

Table 1: Screening Procedural Outline (IM011065)

| Procedure | Screening<br>V1 | Notes |
|---|---|---|
| Eligibility Assessments | | |
| Informed Consent | X | A subject is considered enrolled only when a protocol-specific informed consent is signed. |
| Enroll Subject | X | Obtain number from IRT |
| Inclusion/Exclusion Criteria | X | Includes duration of plaque psoriasis and documentation of presence of plaque psoriasis by the investigator |
| Medical History | X | See Section 5.2 for complete eligibility criteria associated with medical history. Of note, subjects need to be screened for any current uncontrolled neuropsychiatric illness or history of suicidality; any history of TB; any congenital or acquired immunodeficiency; any significant drug allergy such as anaphylaxis; any cancer currently or in the previous 5 years. Investigators are encouraged to check whether subjects have had preventive health measures such as cancer screening (e.g. Pap smear, colonoscopy, mammograms) that is up to date according to local guidelines |
| History of Tobacco Use | X | Include description of current tobacco use. |
| Psoriasis-related History | X | Includes scalp symptoms, PsA/joint pain, nail involvement, palmoplantar involvement, genital involvement, history of other forms of psoriasis. |
| Psoriasis-related Systemic Treatment | X | History of: conventional systemic (eg, methotrexate), biologic, and/or phototherapy. For each therapy, include length of time on treatment and reason(s) for discontinuation (eg, lack of efficacy, intolerance, side effects, loss of access to treatment), if applicable. |
| Other Prior and Concomitant Treatment | X | Includes topical treatments and shampoos for psoriasis and all medications for other conditions such as cardiovascular and mood disorders. |
| Safety Assessments | | |
| Physical Examination | X | Complete PE |
| Physical Measurements | X | Includes height and weight. |
| Vital Signs | X | Includes (ear or oral) body temperature, respiratory rate, seated blood pressure and heart rate. Blood pressure and heart rate should be measured after the subject has been resting quietly for at least 5 minutes. |

Table 1: Screening Procedural Outline (IM011065)

| Procedure | Screening<br>V1 | Notes |
|---|---|---|
| Electrocardiogram | X | ECGs should be recorded after the subject has been supine for at least 5 minutes. |
| Chest Imaging (eg, Chest x-ray) | X | Chest imaging is required if not performed within 6 months of screening visit, copy of radiology report must be on file and reviewed by the investigator. Section 8.4.4. |
| Neuropsychiatric Illness Assessment | X | Based on subject/family response, medical history/medical records, investigator judgment |
| PHQ-8 | X | For establishing baseline depression severity |
| Suicidal Ideation and Behavior Assessment | X | Based on subject/family response, medical history/medical records, investigator judgment |
| eC-SSRS | X | eC-SSRS Assessment: Response of "Actual Suicide Attempt-Lifetime" or suicidal ideation (Severity of 4 or 5) or suicidal behavior will be exclusionary. Rescreening will not be allowed. Section 8.4.7 |
| Monitor for SAEs | X | All SAEs must be collected from the date of subject's written consent until 30 days post discontinuation of dosing or subject's participation in the study. |
| <b>Laboratory Tests</b> | | |
| Hematology | X | Complete Blood Count (CBC) with differential |
| Chemistry Panel | X | |
| Fasting Lipid Panel | X | Subjects are required to fast for at least 10 hours prior to collection. |
| Urinalysis | X | |
| Hemoglobin A1C | X | |
| TSH | X | If TSH above normal reference range, test free T4; if TSH below normal range, test free T4 & T3 |
| hs-CRP | X | |
| Serology | X | Includes HCV antibody, HBsAg, HBsAb, HBcAb, HBV DNA, and HIV antibodies. |
| TB Test | X | In accordance with QuantiFERON-TB (details described in Section 8.4.4). |

Table 1: Screening Procedural Outline (IM011065)

| Procedure | Screening<br>V1 | Notes |
|---|---|---|
| Pregnancy Test (serum) | X | For WOCBP only |
| FSH | X | X To confirm menopausal status (see APPENDIX 4) |
| Clinical Efficacy/Health Outcomes | | |
| sPGA | X | |
| PASI | X | |
| BSA | X | |
| PASE Questionnaire | X | For subjects with peripheral joint complaints to screen for presence of psoriatic arthritis |
| PSSD | X | All consented subjects will be given a diary device at the Screening Visit and will begin recording psoriasis signs and symptoms on a daily basis in the diary device. Subjects who are not randomized will stop recording and return their diary device to the site. Subjects who are randomized will continue recording their psoriasis signs and symptoms on a daily basis in the diary device through Week 52. |

BSA = body surface area; CBC = complete blood count; DNA = deoxyribonucleic acid; ECG = electrocardiogram; eC-SSRS = electronic Columbia Suicide Severity Rating Scale; FSH = follicle stimulating hormone; HBV = hepatitis B virus; HBcAb = hepatitis B core antibody; HBsAb = hepatitis B surface antibody; HBsAg = hepatitis B surface antigen; HCV = hepatitis C virus; HIV = human immunodeficiency virus; hs-CRP = high-sensitivity C-reactive protein; IRT = interactive response technology; PASE = psoriatic arthritis screening and evaluation; PASI = Psoriasis Area and Severity Index; PE = physical examination; PHQ-8 = eight-item Patient Health Questionnaire; PsA = psoriatic arthritis; PSSD = Psoriasis Symptoms and Signs Diary; SAE = serious adverse vent; sPGA = static Physician Global Assessment; T3 = triiodothyronine; T4 = thyroxine; TB = tuberculosis; TSH = thyroid stimulating hormone; V = visit; WOCP = women of childbearing potential.

Table 2: On-Treatment Procedural Outline (IM011065): Week 0 through Week 20

| Procedure | Week 0<br>Baseline / D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Clinical Efficacy/Health<br>Outcomes | | | | | | | | | |
| DLQI | X | X | X | X | X | X | X | | |
| | | | | | | I | | | |
| sPGA | X | X | X | X | X | X | X | | |
| PASI | X | X | X | X | X | X | X | | |
| ss-PGA <sup>a</sup> | X | X | X | X | X | X | | | |
| PGA-F <sup>b</sup> | X | | | X | X | X | | | |
| | | X | X | X | X | X | | | |
| Palmoplantar PGA <sup>c</sup> | X | Λ | Λ | Λ | Λ | Λ | | | |

Table 2: On-Treatment Procedural Outline (IM011065): Week 0 through Week 20

| Procedure | Week 0<br>Baseline / D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|
| PSSD | | | | | | | | | |
| Safety Assessments | | | | | | | | | |
| Complete PE | X | | | | | | X | | |
| Targeted PE | | X | X | X | X | X | | X | See Section 8.4.1 |
| Body Weight | X | | | | | | X | | |
| Vital Signs | X | X | X | X | X | X | X | X | |
| ECG | X | | | | | | X | | |
| PHQ-8 | X | | | | X | | X | | See Section 8.4.6.1 |
| eC-SSRS Assessment | X | | | | X | | X | | Suicidal Ideation and<br>Behavior since last<br>visit |
| Adverse Event Assessment | X | X | X | X | X | X | X | X | |
| Concomitant Medication Use | X | X | X | X | X | X | X | X | |
| <b>Laboratory Tests</b> | | | | | | | | | |
| Hematology | X | X | X | X | X | X | X | X | |
| Lymphocytes Subsets (TBNK) | X | | | | X | | X | | |
| Chemistry Panel | X | X | Х | X | X | X | X | X | If CK >2.5 × ULN,<br>reflex testing is<br>required (see<br>Section 8.4.5) |
| Hemoglobin A1C | X | | _ | | | | X | | |
| hs-CRP | X | X | X | X | X | | X | X | |

Table 2: On-Treatment Procedural Outline (IM011065): Week 0 through Week 20

| Procedure | Week 0<br>Baseline / D1<br>V2 | Week 1<br>D8<br>(±3 d)<br>V3 | Week 2<br>D15<br>(±3 d)<br>V4 | Week 4<br>D29<br>(±3 d)<br>V5 | Week 8<br>D57<br>(±3 d)<br>V6 | Week 12<br>D85<br>(±3 d)<br>V7 | Week 16<br>D113<br>(±3 d)<br>V8 | Week 20<br>D141<br>(±3 d)<br>V9 | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Fasting Lipid Panel | X | | | | X | | X | | Subjects are required<br>to fast for at least 10<br>hours prior to<br>collection |
| Fasting Plasma Glucose | X | | | | X | | X | | |
| Urinalysis | X | | | | | | X | | |
| Serum Immunoglobulin Levels (IgM, IgG, IgA, IgE) | X | | | | X | | X | | |
| Pregnancy Test (Urine) | X | | | X | X | X | X | X | WOCBP Only |
| Study Treatment | | | | | | | | | |
| Randomize | X | | | | | | | | |
| Dispense Study Treatment | X | | X | X | X | X | X | X | |
| Study Treatment Compliance | | X | X | X | X | X | X | X | See Section 6.6 |

CK = creatine kinase: D = Day; d = days: DLOI = Dermatology Life Ouality Index: ECG = electrocardiogram: eC-SSRS = electronic Columbia Suicide
Severity Rating Scale;

C-reactive protein; Ig = immunoglobulin;

PASI = Psoriasis Area and Severity Index: PE = physical examination; PGA =
Physician's Global Assessment: PGA-F = Physician Global Assessment-Fingernails: PHO-8 = eight-item Patient Health Questionnaire;

Symptoms and Signs Diary;

sPGA = static Physician Global Assessment; ss-PGA = scalpspecific Physician's Global Assessment; TBNK = T, B, and natural killer cells;

Wk = Week; WOCP = women of childbearing potential.

Note: All visits  $\pm 3$  Days

<sup>&</sup>lt;sup>a</sup> In subjects with scalp psoriasis at baseline

b In subjects with nail psoriasis at baseline

Clinical Protocol
BMS-986165

IM011065
TYK2 Inhibitor

When multiple assessments are conducted at a single visit, the following is the order in which they should be done:

- 1) Health outcomes assessments
- 2) Safety assessments
- 3) Clinical efficacy assessments
- 4) Laboratory tests (eg, safety laboratory tests,

On fasting days, safety assessments can be done first followed by blood draws, and then health outcomes and, finally, efficacy assessments. The dose of the drug on a visit day is to be taken after blood draws.

c In subjects with palmoplantar psoriasis at baseline

Table 3: On-Treatment Procedural Outline (IM011065): Week 24 through Week 52

| | | | | | / | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup> (or early DC) D365 (±3 d) V17 | Safety<br>Follow-up <sup>b</sup><br>(Week 56)<br>D393<br>(±3 d)<br>V18 | Notes |

Table 3: On-Treatment Procedural Outline (IM011065): Week 24 through Week 52

| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup> (or early DC) D365 (±3 d) V17 | Safety Follow-up (Week 56) D393 (±3 d) V18 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Safety Assessments | | | | | | | | | | |
| Full PE | X | | | | | | | X | X | |
| Targeted Physical<br>Examination | | X | X | X | X | X | X | | | |
| Body Weight | | | | | | | | X | X | |
| Vital Signs | X | X | X | X | X | X | X | X | X | |
| ECG | X | | | | | | | X | | |
| PHQ-8 | | X | | | X | | | X | | See<br>Section 8.4.6.1 |
| eC-SSRS | | X | | | X | | | X | | Suicidal Ideation<br>and Behavior<br>since last visit |
| Adverse Event<br>Assessment | X | X | X | X | X | X | X | X | X | |

Table 3: On-Treatment Procedural Outline (IM011065): Week 24 through Week 52

| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup> (or early DC) D365 (±3 d) V17 | Safety Follow-up (Week 56) D393 (±3 d) V18 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Concomitant<br>Medication Use | X | X | X | X | X | X | X | X | X | |
| <b>Laboratory Tests</b> | | | | | | | | | | |
| Hematology | X | X | X | X | X | X | X | X | X | |
| Lymphocytes Subsets (TBNK) | | | | X | | | | X | | |
| Chemistry Panel | X | X | X | X | X | X | X | X | X | If CPK >2.5 ×<br>ULN, reflex<br>testing is<br>required (see<br>Section 8.4.5) |
| Fasting Lipid Panel | X | | | | | | | X | | Subjects are required to fast for at least 10 hours prior to collection |
| Fasting Plasma<br>Glucose | X | | | | | | | X | | |
| hs-CRP | X | | | X | | | | X | | |
| Hemoglobin A1C | | | | X | | | | X | | |
| Urinalysis | | | | X | | | | X | X | |
| Serum<br>Immunoglobulin<br>Levels (IgM, IgG, IgA,<br>IgE) | | | | X | | | | X | | |

Table 3: On-Treatment Procedural Outline (IM011065): Week 24 through Week 52

| Procedure | Week 24<br>D169<br>(±3 d)<br>V10 | Week 28<br>D197<br>(±3 d)<br>V11 | Week 32<br>D225<br>(±3 d)<br>V12 | Week 36<br>D253<br>(±3 d)<br>V13 | Week 40<br>D281<br>(±3 d)<br>V14 | Week 44<br>D309<br>(±3 d)<br>V15 | Week 48<br>D337<br>(±3 d)<br>V16 | Week 52 <sup>a</sup> (or early DC) D365 (±3 d) V17 | Safety Follow-up (Week 56) D393 (±3 d) V18 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Pregnancy Test (Urine) | X | X | X | X | X | X | X | X | X | WOCBP Only |
| Study Treatment | | | | | | | | | | |
| Dispense Study<br>Treatment | X | X | X | X | X | X | X | | | |
| Study Treatment<br>Compliance | X | X | X | X | X | X | X | X | | |
| BMI = body mass index; eC-SSRS = electronic Columbia-Suicide Severity Rating Scale: CK = creatine kinase: ECG = electrocardiogram; hs-CRP = high-sensitivity C-reactive protein: Ig = immunoglobulin: PE = physical examination: PHO-8 = eight-item Patient Health Ouestionnaire: ULN = upper limit of normal; TBNK = T, B, and natural killer cells; Wk = Week; WOCP = women of childbearing potential | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> For subjects who discontinue from the study prior to Week 52, all Week 52 Visit assessments are to be performed.

When multiple assessments are conducted at a single visit, the following is the order in which they should be done:

- 1) Health outcomes assessments
- 2) Safety assessments
- 3) Clinical efficacy assessments

b For subjects who do not continue in a long-term extension study

4) Laboratory tests (eg, safety laboratory tests,

On fasting days, safety assessments can be done first followed by blood draws, and then health outcomes and, finally, efficacy assessments. The dose of a drug on a visit day is to be taken after blood draws.

### 2 INTRODUCTION

Psoriasis is a chronic inflammatory skin disorder, characterized primarily by erythematous scaly plaques, that affects up to 3% of the general population. Men and women are equally affected and it can present at any age. <sup>1,2</sup> Several studies have observed a bimodal distribution of psoriasis onset with the first peak ranging from 15 to 22 years of age, and the second peak ranging from 55 to 60 years of age. <sup>3,4,5</sup> The most common form of psoriasis (58% to 97% of cases) is plaque psoriasis (psoriasis vulgaris), with less common forms being guttate, pustular, inverse (flexural), and erythrodermic psoriasis. The disease can have a fluctuating relapsing course, with flares that may be induced by factors such as infections, trauma, smoking, and stress.<sup>3</sup> Psoriasis can involve skin in any part of the body; particularly disabling is the involvement of specific anatomic regions, such as hands and feet (palmoplantar), face, scalp and nails. Disease severity can be graded by body surface area (BSA) involvement with mild defined as ≤ 10% BSA, and moderate-to-severe as >10% BSA.<sup>6</sup> Psoriasis has a profound impact on quality of life and can lead to psychological, social and economic consequences, especially in moderate-to-severe disease. This condition is also associated with an increased risk of depression, occurrence of sleep disturbances, social stigma and decreased work productivity. 7,8 Commonly associated comorbidities found in psoriasis patients include diabetes mellitus and metabolic syndrome. In patients with more severe forms of the disease, life expectancy is decreased due to an increase of cardiovascular risk.<sup>9</sup>

Treatments include topical preparations, eg, corticosteroids, vitamin D analogues, calcineurin inhibitors, and salicylic acid; phototherapy modalities, including PUVA (psoralens with UVA) and narrow band UVB; and systemic therapies. In moderate-to-severe disease, systemic treatments are usually needed and may include oral agents (retinoids, methotrexate, cyclosporine, and apremilast) or injectables (eg, biologics such as tumor necrosis factor (TNF) inhibitors etanercept, infliximab, and adalimumab) anti-IL-12/23p40 antibody (ustekinumab), IL-17 antagonists (secukinumab, ixekizumab, and brodalumab), and anti-IL-23p19 antibody (guselkumab). Many of these treatments are associated with increased risk of adverse events (AEs) such as hepatotoxicity and neutropenia (methotrexate);<sup>10</sup> nephrotoxicity (cyclosporine);<sup>11</sup> depression and weight loss (apremilast);<sup>12</sup> serious infections (cytokine inhibitors);<sup>13,14,15,16</sup> candidiasis and Crohn's disease (IL-17 antagonists).<sup>16, 17, 18</sup>

Although effective therapeutic options are available, under-treatment or nontreatment of psoriasis has been reported in up to half of surveyed patients (based on absence of treatment and/or dissatisfaction with treatment). Many patients with severe disease are still being managed with only topicals, and many patients consider their psoriasis treatment to be inadequate. Accordingly, there remains a need for more effective oral options, when compared with currently available agents, that would increase adherence to treatment.

### 2.1 Study Rationale

BMS-986165 could be a therapeutic option for the treatment of subjects with moderate-to-severe plaque psoriasis based on results of a recently completed 12-week, randomized, Phase 2, placebo-controlled, parallel-group study with 5 different BMS-986165 treatment arms: 3 mg every

other day (QOD); 3 mg once daily (QD); 3 mg twice daily (BID); 6 mg BID; and 12 mg QD (Study IM011011). Overall, 267 subjects were randomized (44 to 45 subjects per treatment arm) in the Phase 2 study. All BMS-986165 treatment groups, except 3 mg QOD, achieved the primary endpoint of superiority compared with placebo in the proportion of subjects achieving PASI 75 after 12 weeks of treatment. Compared with placebo treatment group, in which 6.7% of the subjects achieved PASI 75 response, 38.6% (P = 0.0003), 68.9% (P < 0.0001), 66.7% (P < 0.0001) and 75% (P < 0.0001) of subjects treated with 3 mg QD, 3 mg BID, 6 mg BID, and 12 mg QD achieved PASI 75, respectively. The PASI 75 responses plateaued at a dose of 3 mg BID. Also, there was a clinically significant proportion of subjects treated with BMS-986165 achieving an sPGA score of 0 or 1 compared with placebo at Week 12. Compared with the placebo treatment group in which 6.7% of the subjects achieved an sPGA score of 0 or 1, 41.5%, 75.6%, 65.9%, and 75% of the subjects treated with 3 mg QD, 3 mg BID, 6 mg BID, and 12 mg QD achieved an sPGA score of 0 or 1, respectively with responses again plateauing at dose of 3 mg BID. The Phase 3 dose selected (6 mg QD) is expected to demonstrate equivalent efficacy to the 3 mg BID dose.

This Phase 3 study is designed to confirm the efficacy and safety of BMS-986165 6 mg QD in a population of subjects with moderate-to-severe plaque psoriasis.

# 2.2 Background

Tyrosine kinase 2 (TYK2) is a nonreceptor tyrosine kinase associated with receptors for the p40-containing cytokines IL-12 and IL 23, as well as the Type I interferon (IFN) receptor, and is required for the activation of their downstream signaling pathways. TYK2 catalyzes the phosphorylation of the intracellular receptor domains and signal transducer and activator of transcription (STAT) proteins resulting in the activation of STAT-dependent transcription and functional responses specific for these cytokines. <sup>20,21,22</sup> Because TYK2-dependent cytokines (eg, Type I IFNs, IL-12, IL-23) are distinct from those dependent on closely related Janus kinase (JAK) family members JAK1/JAK3 (eg, IL-2, IL-15, IL-7) or JAK2 (eg, erythropoietin, thrombopoietin, GM-CSF), a TYK2 inhibitor would be expected to have a highly differentiated profile from inhibitors of other JAK family kinases. TYK2 dependent pathways and the cytokine networks they modulate (eg, IL-23/IL-17, IFNα) have been implicated in the pathophysiology of multiple immune-mediated diseases, including psoriasis, lupus, spondyloarthritides, and Crohn's disease.

BMS-986165 is a potent, highly selective, oral small molecule inhibitor of TYK2. A comprehensive in vitro and in vivo characterization of BMS-986165 has been established and supports the development of this compound in humans. Inhibition of TYK2 is expected to provide therapeutic benefit for subjects with psoriasis for multiple reasons: 1) Many of the pathways in the TYK2 signaling cascade (IL-23 and the downstream mediators IL-17 and IL-22; IFNα) have been implicated in pathogenesis of psoriasis. <sup>7</sup> 2) Biologic agents targeting the IL-17, IL-23p19, and IL-12/23 p40 pathways have been approved for and are highly efficacious in the treatment of psoriasis.

# 2.2.1 Early Clinical Development

The clinical data available to date supporting the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of BMS-986165 are from 5 completed Phase 1 studies in healthy subjects (IM011002, IM011015, IM011016, IM011031, and IM011039) and 1 completed Phase 2 study in adult subjects with moderate-to-severe plaque psoriasis (IM011011).

Overall, BMS-986165 has been generally well tolerated across all studies, and no safety issues have been identified to limit the investigation of the dose of BMS-986165 up to 12 mg QD in further clinical studies. A detailed description of the chemistry, pharmacology, efficacy, and safety of BMS-986165 is provided in the Investigator Brochure (IB).





# 3 OBJECTIVES AND ENDPOINTS

Table 4: Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| Assess whether BMS-986165 is superior to placebo at Week 16 in the treatment of subjects with moderate-to-severe plaque psoriasis | static Physician Global Assessment (sPGA) 0/1 response Psoriasis Area and Severity Index (PASI) 75 response (defined as a 75% improvement in PASI score from baseline) |
| Secondary | |
| Assess whether BMS-986165 is superior to placebo over<br>the first 16 weeks of treatment | • sPGA 0/1 response |
| | PASI 90 response |
| | sPGA 0 response |
| | PASI 100 response |
| Assess whether BMS-986165 is superior to placebo in nail | • PGA-F 0/1 |
| psoriasis through Week 16 in those subjects who have baseline Physician's Global Assessment of Fingernail Psoriasis (PGA-F) score ≥3 | |
| Assess whether BMS-986165 is superior to placebo in palmoplantar psoriasis through Week 16 in those subjects who have baseline palmoplantar Physician's Global Assessment (pp-PGA) score ≥3 | • pp-PGA 0/1 response |

Table 4: Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Evaluate improvement in patient reported outcomes for<br>BMS-986165 compared with placebo through Week 16 | Change from baseline in Psoriasis Symptoms and Signs Diary (PSSD) symptom score |
| | • PSSD symptom score of 0 (among subjects with a baseline PSSD symptom score ≥1) |
| | • DLQI 0/1 (among subjects with a baseline DLQI score ≥2) |

# 4 STUDY DESIGN

# 4.1 Overall Design

Study IM011065 will be a 52-week, multi-center, randomized double-blind, placebo-controlled study to evaluate the safety and efficacy of BMS-986165 vs placebo. A total of approximately 219 qualified subjects with moderate-to-severe plaque psoriasis in mainland China, Taiwan, and

South Korea will be enrolled (see additional details in Section 4.2).

The duration of study participation is approximately 60 weeks, and will be divided into the following periods: screening (up to 4 weeks), treatment (52 weeks), and follow-up (4 weeks).

Physical exams, 12-lead ECGs, and clinical laboratory evaluations will be done at select visits during the study. Subjects in this study will be monitored for AEs.

### 4.1.1 Screening Period

Subjects will be evaluated during the screening period to ensure that they meet eligibility criteria. A detailed medical history will be done at this time, as well as a complete physical exam. Psoriasis-related history, which will include length of diagnosis, body involvement, and history of systemic treatment, will be assessed here. Depression and suicidality assessments will also be performed. An evaluation for tuberculosis will be done based on medical history, recent chest imaging, and a QuantiFERON-TB test.

### 4.1.2 Treatment Period

Qualified subjects who have completed the screening procedures and have met the inclusion/exclusion criteria will be randomized on Day 1 in a 2:1 ratio to either BMS-986165 6 mg QD or placebo, respectively.

Dummy tablets (placebo to BMS-986165 6 mg tablets) will be administered to subjects to maintain blinding. Additional details are provided in Section 6.1.

Randomization should not occur until at least 8 days after the screening visit to allow collection of PSSD data during screening in order to calculate a baseline PSSD score. Randomization will be stratified by country (mainland China vs. non-mainland China) and previous biologic use (for psoriasis, psoriatic arthritis or other inflammatory diseases only; yes/no).

### 4.1.3 Week 16

The coprimary endpoints (sPGA 0/1 and PASI 75) will be assessed at Week 16. Subjects receiving placebo will be switched in a blinded manner to BMS-986165 6 mg QD at Week 16. Subjects who are randomized to BMS-986165 6 mg QD will continue their treatment regimen through Week 52.

#### 4.1.4 Week 24

At Week 24, a subject who has may be treated with restricted topicals/shampoos as described in Section 6.7.1 at the investigator's discretion. These treatments may be initiated only at Week 24 and not at subsequent time points. A subject who is started on these treatments at Week 24 may use them as needed per the investigator's judgement through Week 52.

# 4.1.5 Week 52 and Follow-up Period

The follow-up period is a 4-week window after the Week 52 visit, unless the subject rolls over into the long-term extension. The subject will be encouraged to report any SAEs or AEs experienced during this time.

Subjects who discontinue study treatment early should remain in the study for protocol-specified procedures (please refer to Section 7.1 for more details).

Subjects completing 52 weeks of treatment will be offered the opportunity to roll over to a separate long-term extension study ( $\geq 2$  years) where they will be treated with BMS-986165 6 mg QD.

The study design schematic is presented in Figure 1.

Figure 1: Study Design Schematic



QD = once daily.

The coprimary endpoints will be evaluated at Week 16.

### 4.1.6 Data Monitoring Committee and Other External Committees

# 4.1.6.1 Data Monitoring Committee

An external data monitoring committee (DMC) with multi-disciplinary representation will be established to evaluate on a periodic basis; AEs, laboratory measurements, and safety assessments to ensure the ongoing safety of study subjects. An independent reporting statistician not involved in the conduct of the study will be designated by to provide the DMC with essential safety data during the study.

The DMC responsibilities, authorities, and procedures will be documented and followed according to the DMC charter.

### 4.1.6.2 Infection Adjudication Committee

An independent Infection Adjudication Committee, composed of individuals with relevant expertise, will review in a blinded manner and adjudicate infection AEs, such as opportunistic infections, influenza, herpes zoster, and TB, reported in the study per criteria specified in a separate charter. Additional information about these infections may be collected on the case report form in order to characterize and understand them. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee is distinct from the DMC and Adjudication Committee members will not be investigators on the study.

# 4.1.6.3 CV Adjudication Committee

An independent cardiovascular (CV) Adjudication Committee, composed of individuals with relevant expertise, will review in a blinded manner and adjudicate cardiovascular and cerebrovascular AEs such as, but not limited to, Major Adverse Cardiovascular Events (MACE) that include death, non-fatal myocardial infarction, non-fatal stroke; revascularization procedures; heart failure; dysrhythmias; heart blocks; and thrombotic events reported in the study per criteria specified in a separate charter. Additional information about cardiovascular and cerebrovascular AEs may be collected on the case report form in order to characterize and understand them. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee is distinct from the DMC and Adjudication Committee members will not be investigators on the study.

### 4.1.6.4 Suicidal Ideation and Behavior Adjudication Committee

An independent Suicidal Ideation and Behavior Adjudication Committee, composed of individuals with relevant expertise, will review in a blinded manner and adjudicate suicidal ideation/behavior reported in the study per criteria specified in a separate charter. Additional information about suicidal ideation/behavior may be collected on the case report form. The Adjudication Committee members will be blinded to the treatment assignment of subjects. The structure, responsibilities, and procedures of the Adjudication Committee will be outlined in a charter. The Adjudication Committee is distinct from the DMC and Adjudication Committee members will not be investigators on the study.

# 4.2 Number of Subjects

Approximately 219 qualified subjects will be randomized in a 2:1 ratio to BMS-986165 6 mg QD or placebo, respectively.

### 4.3 End of Study Definition

The duration of study participation for individual subjects is expected to be up to 60 weeks (420 days), which includes screening (up to 4 weeks), treatment (52 weeks) and follow-up (up to 4 weeks) periods.

The start of the study is defined as first visit for first subject screened. The end of the study is defined as the last visit or scheduled procedure shown in the Schedule of Activities (Section 1.3) for the last subject. Study completion is defined as the final date on which data was or is expected to be collected (Week 56 for collection of potential SAEs).

# 4.4 Scientific Rationale for Study Design

This Phase 3 study will be conducted in a population of subjects with stable moderate-to-severe plaque psoriasis who are candidates for systemic psoriasis therapy. The study is designed to confirm the efficacy and safety of BMS-986165 compared with placebo in achieving sPGA of 0/1 and PASI 75 at Week 16. The sPGA and PASI 75 are standard measures in clinical trials of demonstrating efficacy of systemic psoriasis treatments. The placebo arm is included in this study for a duration of 16 weeks to provide a control for the natural fluctuation of psoriasis activity that may occur and to provide a safety standard for comparison. Subjects in the placebo arm will be switched to BMS-986165 at Week 16 to provide them psoriasis treatment after the coprimary endpoints are collected.



#### 5 STUDY POPULATION

Eligibility criteria for this study have been carefully considered to ensure 1) selection of appropriate subjects with psoriasis, 2) safety of the study subjects and 3) the results of the study can be used for regulatory filing and other purposes. It is imperative that subjects fully meet all eligibility criteria.

All screening and randomization evaluations must be completed and reviewed to confirm that potential subjects meet all eligibility criteria. The investigator will maintain a screening log to record details of all subjects screened and to confirm eligibility or record reasons for screening failure, as applicable.

### 5.1 Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

### 1) Signed Written Informed Consent

a) Subjects must be willing to participate in the study and sign the informed consent form (ICF)

# 2) Type of Subject and Target Disease Characteristics

- a) N/A
- b) Deemed by the investigator to be eligible for phototherapy or systemic therapy
- c) ≥10% of BSA involvement at screening visit and Day 1
- d) Psoriasis Area and Severity Index (PASI) score ≥12 and static Physician's Global Assessment (sPGA) ≥3 at screening visit and Day 1
- e) Men and women in mainland China, Taiwan, and South Korea diagnosed with stable plaque psoriasis for 6 months or more. Stable psoriasis is defined as no morphology changes or significant flares of disease activity in the opinion of the investigator

### 3) Age and Reproductive Status

- a) Men and women aged ≥18 years or legal age at the time of screening visit
- b) Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening visit, and a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug
- c) Women must not be pregnant, lactating, breastfeeding or planning pregnancy during the study period
- d) Women of childbearing potential must agree to use correctly a highly effective method(s) of contraception for the duration of treatment (52 weeks) with study drug(s) BMS-986165 plus 5 half-lives of study drug (3 days) plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion (total of 33 days after last dose of study drug). WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements, but must still undergo pregnancy testing as described in this protocol
- e) Male subjects who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (APPENDIX 4 for the duration of treatment with study
Clinical Protocol BMS-986165

treatment(s) plus 5 half-lives of the study treatment (3 days) for a total of 3 days post-treatment completion. In addition, male subjects must be willing to refrain from sperm donation during this time

Investigators shall counsel WOCBP, and male subjects who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, (APPENDIX 4) which have a failure rate of < 1% when used consistently and correctly.

#### 5.2 Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

### 1) Target Disease Exceptions

a) Has nonplaque psoriasis (ie, guttate, inverse, pustular, erythrodermic or drug-induced psoriasis) at screening or Day 1

### 2) Infectious/Immune-related Exclusions

- a) History or evidence of outpatient active infection and/or febrile illness within 7 days prior to Day 1
- b) History of serious bacterial, fungal, or viral infection requiring hospitalization and/or intravenous (IV) antimicrobial treatment within 60 days prior to Day 1
- c) Any untreated bacterial infection within 60 days prior to Day 1
- d) Any ongoing evidence of chronic, bacterial infection (eg, chronic pyelonephritis, chronic osteomyelitis, chronic bronchiectasis)
- e) Any history of proven infection of a joint prosthesis in which the prosthesis was not removed or replaced, or received antibiotics for suspected infection of a joint prosthesis in which the prosthesis was not removed or replaced
- f) Received live vaccines within 60 days prior to Day 1, or plans to receive a live vaccine during the study, or within 60 days after completing study treatment
- g) Presence of herpes zoster lesions at screening or Day 1
- h) History of serious herpes zoster or serious herpes simplex infection which includes, but is not limited to, any episode of disseminated herpes simplex, multidermatomal herpes zoster, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (recurrent is defined as 2 episodes within 2 years)
- i) Evidence of, or test positive for, hepatitis B virus (HBV) at Screening. Positive hepatitis B lab testing is defined as: 1) Positive hepatitis B surface antigen (HBsAg+) **OR** 2) Presence of hepatitis B virus deoxyribonucleic acid (DNA) **OR** 3) Positive anti-hepatitis B core antibody without concurrent positive hepatitis B surface antibody (HBcAb+ and HBsAb-)
- j) Evidence of, or test positive for, hepatitis C virus (HCV) at screening. A positive test for HCV is defined as: 1) positive for hepatitis C antibody (anti-HCVAb) **AND** 2) positive via a confirmatory test for HCV (eg, HCV polymerase chain reaction)

- k) Positive for human immunodeficiency virus by antibody testing (HIV-1 and -2 Ab) at screening
- l) Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the subject's immune status (eg, history of opportunistic infections [eg, *Pneumocystis jirovecii* pneumonia, histoplasmosis, or coccidioidomycosis], history of splenectomy, primary immunodeficiency)

### 3) Any of the following tuberculosis (TB) criteria:

- a) History of active TB prior to screening visit, regardless of completion of adequate treatment
- b) Signs or symptoms of active TB (eg, fever, cough, night sweats, and weight loss) during screening as judged by the investigator
- c) Any imaging of the chest (eg, chest x-ray, chest computed tomography [CT] scan) obtained during the screening period or anytime within 6 months prior to screening with documentation, showing evidence of current active or history of active pulmonary TB
- d) Latent TB infection (LTBI) defined as positive IFN gamma release assay (IGRA), by QuantiFERON-TB testing at screening, in the absence of clinical manifestations
  - Note: Subject is eligible if (i) there are no current signs or symptoms of active TB AND (ii) subject has received adequate documented treatment for LTBI within 5 years of screening **OR** has initiated prophylactic treatment for LTBI per local guidelines and is rescreened after 1 month of treatment. To continue in the study, subject must agree to complete a locally-recommended course of treatment for LTBI.

Note: An IGRA test that is indeterminate with no signs or symptoms of active TB must be re-tested for confirmation. If the second test is again indeterminate the subject will be excluded from the study. If the re-test is positive, the subject should be treated as having LTBI. If the re-test is negative, subject may be eligible provided no other exclusion criteria for TB are met.

### 4) Medical History and Concurrent Diseases

- a) Any major surgery within 8 weeks prior to Day 1, or any planned surgery for the first 52 weeks of the study
- b) Has donated blood >500 mL within 4 weeks prior to Day 1, or plans to donate blood during the course of the study
- c) Drug or alcohol abuse, as determined by the investigator, within 6 months prior to Day 1
- d) Medical marijuana or prescription marijuana taken for medicinal reasons
- e) Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, psychiatric, neurologic, immunologic, or local active infection/infectious illness) that, in the investigator's judgment or after consultation with the Medical Monitor, will substantially increase the risk to the subject if he or she participates in the study
- f) Unstable cardiovascular disease, defined as a recent clinical cardiovascular event (eg, unstable angina, myocardial infarction, stroke, rapid atrial fibrillation) in the last 3 months

prior to screening, or a cardiac hospitalization (e.g. revascularization procedure, pacemaker implantation) within 3 months prior to screening

g) Has uncontrolled arterial hypertension characterized by a systolic blood pressure (BP) >160 mm Hg or diastolic BP >100 mm Hg

Note: Determined by 2 consecutive elevated readings. If an initial BP reading exceeds this limit, the BP may be repeated once after the subject has rested sitting for  $\geq 10$  minutes. If the repeat value is less than the criterion limits, the second value may be accepted

- h) Class III or IV congestive heart failure by New York Heart Association Criteria
- i) Has cancer or history of cancer (solid organ or hematologic including myelodysplastic syndrome) or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma, or carcinoma of cervix in situ that has been treated with no evidence of recurrence)
- j) Any significant/uncontrolled neuropsychiatric illness as clinically judged by the investigator during screening or at Day 1

#### **OR**

Any lifetime history of suicidal ideation, suicidal behavior, or suicidal attempts by medical history or by electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) documentation, or by answering "yes" to Question 4 or 5 which indicates a suicidal ideation severity level of 4 or 5 on the eC-SSRS at Screening or at Day 1, or is clinically deemed to have a suicide risk by the investigator

- k) Prior exposure to investigational product (ie, BMS-986165)
- l) If the subject has received biologics previously, the following exclusion criteria for washout will apply:
  - i) Antibodies to IL-12, IL-17 or IL-23 (eg, ustekinumab, secukinumab, tildrakizumab, ixekizumab, or guselkumab) within 6 months of Day 1
  - ii) TNF inhibitor(s) (e.g. etanercept, adalimumab, infliximab, certolizumab) within 2 months of Day 1
  - iii) Agents that modulate integrin pathways to impact lymphocyte trafficking (eg, natalizumab), or agents that modulate B cells or T cells (eg, alemtuzumab, abatacept, or visilizumab) within 3 months of Day 1
  - iv) Rituximab within 6 months of Day 1
- m) Has received systemic non-biologic psoriasis medications and/or any systemic immunosuppressants (including, but not limited to, methotrexate, azathioprine, cyclosporine, JAK inhibitors, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus, oral or injectable corticosteroids, retinoids, 1,25-dihydroxy vitamin D3 and analogues, psoralens, sulfasalazine, or fumaric acid derivatives) within 4 weeks prior to Day 1

- n) Has used leflunomide within 6 months prior to Day 1
- o) Has used opioid analgesics within 4 weeks prior to Day 1
- p) Has received lithium, antimalarials, or intramuscular (IM) gold within 4 weeks of the first administration of any study medication
- q) Has received phototherapy (including either oral and topical PUVA light therapy, ultraviolet B [UVB] or self-treatment with tanning beds or therapeutic sunbathing) within 4 weeks prior to Day 1
- r) Has used topical medications/treatments that could affect psoriasis evaluation (including, but not limited to, high potency corticosteroids (WHO Classes I-V), >3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, pimecrolimus, and tacrolimus) within 2 weeks prior to Day 1
  - Note: Low potency topical steroids (WHO Class VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta-hydroxy acids or other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit.
- s) Use of shampoos that contain corticosteroids, coal tar, >3% salicylic acid, or vitamin D3 analogues within 2 weeks prior to Day 1
- t) Has received an experimental antibody or experimental biologic therapy within the previous 6 months, **OR** received any other experimental therapy or new investigational agent within 30 days or 5 half-lives (whichever is longer) prior to Day 1 **OR** is currently enrolled in an investigational study
- u) Any botanical preparations (eg, herbal supplements or traditional Chinese medicines derived from plants, minerals, or animals) intended to treat psoriasis or other immunological diseases within 4 weeks prior to Study Day 1
- v) Any other sound medical, psychiatric and/or social reasons as determined by the investigator

### 5) Physical and Laboratory Evaluations

- a) At screening
  - i) Absolute WBC count <3000/mm<sup>3</sup>
  - ii) Absolute lymphocyte count <500/mm<sup>3</sup>
  - iii) Absolute neutrophil count <1000/mm<sup>3</sup>
  - iv) Platelet count <100,000/mm<sup>3</sup>
  - v) Hemoglobin < 9 g/dL
  - vi) ALT and/or AST >3X upper limit of normal (ULN)
  - vii) Total, unconjugated, and/or conjugated bilirubin >2 × ULN
  - viii) Thyroid stimulating hormone (TSH) outside the normal range

#### **AND**

Free T4 (thyroxine) or T3 (triiodothyronine) outside the normal reference range

- b) ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the subject if participating in the study
- c) Renal impairment based on an estimated glomerular filtration rate (eGFR) <45 mL/min
- d) Inability to be venipunctured and/or tolerate venous access
- e) Any other significant laboratory abnormalities that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study

### 6) Allergies and Adverse Drug Reactions

a) History of any significant drug allergy (such as anaphylaxis)

### 7) Other Exclusion Criteria

- a) Prisoners or subjects who are involuntarily incarcerated. (Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a subject. Strict conditions apply and BMS approval is required).
- b) Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
- c) Inability to comply with restrictions and prohibited activities/treatments as listed in the study protocol
- d) Site personnel or their immediate family

# 5.3 Lifestyle Restrictions

General skin care measures (with above restrictions for topical treatments) that are standard for patients with plaque psoriasis are permitted. Subjects should avoid excessive sun exposure and avoid risks that are known to provoke flare of psoriasis.

# 5.3.1 Meals and Dietary Restrictions

Study treatment may be taken without regard to meals; however, subjects are required to fast for a minimum of 10 hours before visits on which fasting lipid, fasting glucose samples will be drawn.

## 5.3.2 Caffeine, Alcohol, and Tobacco

No restrictions are required; however, extensive use of caffeine, alcohol and tobacco should be avoided.

# 5.3.3 Activity

No restrictions are required; however, unusual physical exertion should be avoided during the study.

#### 5.4 Screen Failures

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently randomized in the study for any reason. A minimal set of screen failure information is required to ensure transparent reporting of screen failure subjects, to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements, and to respond to queries from regulatory authorities. Minimal set of screen failure information includes date of consent, demography, screen failure details (ie, eligibility criteria that the subject did not meet), and any serious AEs during the screening period.

### 5.4.1 Retesting During Screening or Rescreening

For laboratory parameters that initially do not meet eligibility requirements, a single retest within the 28-day screening period is permitted before subject is declared a screen failure. This is an effort to find all possible well-qualified subjects. Consultation with the medical monitor may be needed to identify whether repeat testing of any particular parameter would be clinically relevant.

The study permits the rescreening (after the end of the initial 28-day screening period) of a subject who discontinues the study as a pretreatment failure (ie, the subject fails to meet eligibility criteria and has not been treated). The subject must be reconsented, will be assigned a new identification number, and a full screening visit must be performed again. A subject can only be rescreened 1 time (ie, if the subject fails 1 rescreening attempt, no additional rescreening is allowed). Depending on the timing of rescreening, repeat chest imaging may not be required. Duration of existing treatments and required discontinuation periods shall be considered relative to the new screening visit and/or randomization.

The most current result prior to randomization is the value by which study inclusion will be assessed, as it represents the subject's most current clinical state.

### 6 TREATMENT

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo, or medical device intended to be administered to a study subject according to the study randomization or treatment allocation.

Study treatment includes both Investigational [Medicinal] Product (IP/IMP) and Non-investigational [Medicinal] Product (Non-IP/Non-IMP) and can consist of the following: BMS-986165 and placebo.

An IP, also known as IMP in some regions, is defined a pharmaceutical form of an active substance or placebo being tested or used as a reference in a clinical study, including products already with a marketing authorization but used or assembled (formulated or packaged) differently than the authorized form, or used for an unauthorized indication, or when used to gain further information about the authorized form.

Other medications used as support or escape medication for preventative, diagnostic, or therapeutic reasons, as components of the standard of care for a given diagnosis, may be considered as non-IP. Table 5 shows the study treatments for Protocol IM011065.

Table 5: Study Treatments for IM011065

| Product<br>Description /<br>Class and<br>Dosage Form | Potency | IP/Non-IP | Blinded or<br>Open Label | Packaging /<br>Appearance | Storage<br>Conditions<br>(per label) |
|---|---|---|---|---|---|
| BMS-986165<br>tablet | 6 mg | IP | Blinded | Bottle | Store 15°C to<br>25°C; Store in a<br>tightly closed<br>container;<br>Protect from<br>light |
| Placebo tablet<br>to match<br>BMS-986165<br>6 mg | n/a | IP | Blinded | Bottle | Store 15°C to<br>25°C; Store in a<br>tightly closed<br>container;<br>Protect from<br>light |

IP = investigational product; n/a = not applicable

### 6.1 Treatments Administered

Study treatment will be administered as described in Section 4.1.2. The selection and timing of dose for each subject is as follows:

Table 6: Selection and Timing of Dose

| Study Treatment | Unit dose<br>strength(s)/Dosage<br>level(s) | Dosage formulation<br>Frequency of Administration | Route of<br>Administration |
|---|---|---|---|
| BMS-986165 | 6 mg | 1 active tablet QD in the morning | oral |
| Placebo QD | n/a | 1 BMS-986165 placebo QD in the morning | oral |

 $\overline{QD}$  = once daily, n/a = not applicable

# 6.2 Method of Treatment Assignment

Before the study is initiated, each user (at investigative sites) will receive log-in information and directions on how to access the interactive response technology (IRT) system. At the time of the screening visit, immediately after informed consent is obtained and before any study-related procedures are performed, the investigative site will access the enrollment option of the IRT system for assignment of a subject number for all subjects, including subjects not subsequently randomized or treated. The subject number is assigned sequentially by the system and will be unique across all sites. All enrolled subjects will be assigned sequential subject numbers. The subject number will not be used for any other subject. If a subject is rescreened, they will be given a new identification number.

At Week 0 (Day 1), subjects who meet all criteria for enrollment at Screening and Day 1 will be centrally randomized in a 2:1 ratio to BMS-986165 6 mg QD or placebo as determined by a computer-generated randomization schedule using IRT. The randomization lists will be generated by the IRT vendor using a permuted block design within each stratum level. The randomization in this study will be stratified by country (mainland China vs. non-mainland China) and previous biologic use for psoriasis, psoriatic arthritis or other inflammatory diseases only (yes/no). After all inclusion/exclusion criteria have been met for a subject, the investigative site will access the IRT on Day 1 for the purpose of randomizing a subject. A treatment group will be assigned by IRT based on the above-described randomization schedule and each subject will be assigned a unique randomization number. In addition, a unique kit number will be assigned to the subject corresponding to the treatment assignment.

A kit will contain adequate study treatment for a 4-week supply. At subsequent visits, when new treatment kits need to be provided, the investigative site will access the IRT to obtain the kit number to assign to the subject. Study treatment will be dispensed at study visits as shown in the Schedule of Activities (Section 1.3).

At Week 16, subjects receiving placebo will be switched in a blinded manner to BMS-986165 6 mg QD.

### 6.3 Blinding

### 6.3.1 Maintaining the Blind

Blinded treatment assignments will be managed using IRT. IP supply will be controlled by IRT at each visit.

All tablets are identical in appearance and will be supplied in bottles with each daily dose made up of the appropriate combination of active and/or placebo tablets to provide the correct treatment, as shown in Table 5. Investigative site staff, Sponsor and designee personnel, and subjects and their families will remain blinded to treatment assignments.



# 6.3.2 Circumstances for Unblinding

Blinding of treatment assignment is critical to the integrity of this clinical study. However, in the event of a medical emergency or pregnancy in an individual subject in which knowledge of the IP is critical to the subject's management, the blind for that subject may be broken by the investigator. The subject's safety takes priority over any other considerations in determining if a treatment assignment should be unblinded.

Before breaking the blind of an individual subject's treatment, the investigator should determine that the unblinded information is necessary, ie, that it will alter the subject's immediate

management. In many cases, particularly when the emergency is clearly not related to the IP, the problem may be properly managed by assuming that the subject is receiving active product. It is highly desirable that the decision to unblind treatment assignment be discussed with the medical monitor, but the investigator always has ultimate authority for the decision to unblind. The Principal Investigator should only call in for emergency unblinding AFTER the decision to discontinue the subject has been made.

In case of an emergency, the investigator has unrestricted access to randomization information via IRT and is capable of breaking the blind through the IRT system without prior approval from the sponsor. After the unblinding, the investigator shall notify the medical monitor and/or study director. The method of unblinding for emergency purposes is described in the IRT manual. Subject and unblinded treatment information and the reason for the blind being broken must be recorded on the appropriate study status page of the electronic case report form (eCRF). After unblinding via IRT, the investigator shall notify the Medical Monitor.

In cases of accidental unblinding, contact the Medical Monitor and ensure every attempt is made to preserve the blind. Any request to unblind a subject for non-emergency purposes must be discussed with the Medical Monitor prior to unblinding.

If a subject is unblinded for any reason, the subject will be discontinued from treatment.

### 6.3.3 Unblinding for Week 16 Primary Endpoint Analysis

An unblinded analysis of data through Week 16 will be performed after all subjects complete their Week 16 visit or have discontinued prior to Week 16. A select group of personnel who are not involved in the conduct of the study will review the results to write a clinical study report. Following the Week 16 analysis until the end of the study, the investigators, subjects, and clinical trial team members who directly cooperate with the site staff will continue to remain blinded to the initial treatment assignment. Details of maintaining the blind following the unblinded analysis will be finalized prior to the Week 16 database lock. A final analysis will be performed after all subjects complete the Week 52 visit or discontinue prior to the Week 52 visit, and a clinical study report will be written.

### 6.4 Dosage Modification

There is no provision for dose modification of study treatment. If a subject interrupts treatment due to an AE, study treatment can be restarted in consultation with the Medical Monitor.

# 6.5 Preparation/Handling/Storage/Accountability

The IP should be stored in a secure area according to local regulations. It is the responsibility of the investigator to ensure that the IP is only dispensed to study subjects. The IP must be dispensed only from official study sites by authorized personnel according to local regulations.

The product storage manager should ensure that the study treatment is stored in accordance with the environmental conditions (temperature, light, and humidity) as determined by BMS. If concerns regarding the quality or appearance of the study treatment arise, the study treatment should not be dispensed and BMS should be contacted immediately.

Investigational product documentation (whether supplied by BMS or not) must be maintained that includes all processes required to ensure drug is accurately administered. This includes documentation of drug storage, administration and, as applicable, storage temperatures, reconstitution, and use of required processes (eg, required diluents, administration sets).

• Guidance and information for final disposition of unused study treatment are provided in APPENDIX 2.

### 6.5.1 Retained Samples for Bioavailability/Bioequivalence

Not applicable.

### 6.6 Treatment Compliance

Study treatment compliance will be periodically monitored using standard drug accountability procedures (comparing the number of tablets returned to number dispensed, considering the expected regimen and any reported missed doses). Drug accountability will be reviewed by the investigative site staff at each visit to confirm treatment compliance. Site staff will discuss any discrepancies with the subject and remind the subject of the importance of compliance with the assigned regimen. A real-time monitoring platform may be used.

### 6.7 Concomitant Therapy

### 6.7.1 Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications in the study are described below. Medications taken within 4 weeks prior to study drug administration must be recorded on the CRF.

- 1) Exposure to any investigational drug or placebo outside of the current study
- 2) Use of any medications/therapy that would aggravate psoriasis. These include agents such as lithium, antimalarials (quinacrine, chloroquine, and hydroxychloroquine), propranolol, indomethacin, and quinidine unless it is considered necessary for the subject's welfare and/or treatment of an AE/SAE
- 3) Use of opioid analgesics unless it is considered necessary for the subject's welfare and / or treatment of an AE/SAE
- 4) Phototherapy; use of tanning booths or therapeutic sunbathing
- 5) Any use of biologic medications (eg. adalimumab, etanercept, infliximab, ustekinumab)
- 6) Any use of oral psoriasis medications (eg, methotrexate, cyclosporine, retinoids, fumaric acid derivatives) for any indication
- 7) Any use of oral or injectable corticosteroids (prednisone, methylprednisolone, etc.), unless it is considered necessary for the subject's welfare and/or treatment of an AE/SAE
- 8) Note: otic, ophthalmic, nasal, or inhaled corticosteroids within recommended doses and with no systemic effects are permitted.
- 9) Any topical medications/treatments, which are used for any indication, that could affect psoriasis evaluation (including, but not limited to, high potency corticosteroids [WHO Classes I-V], >3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene,

vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, pimecrolimus, and tacrolimus)

Exception: The following topical treatments may be initiated only at Week 24 per investigator's discretion in subjects who have (see Section 4.1.4)

• High potency corticosteroids (WHO Classes I-V), >3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene, vitamin D derivatives, retinoids, tazarotene

Note: Low potency topical steroids (WHO Class VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta-hydroxy acids or other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit.

10) Any medicated shampoos that contain corticosteroids, coal tar, >3% salicylic acid, or vitamin D3 analogues

Exception: The above shampoos may be initiated only at Week 24 per investigator's discretion in subjects who have (see Section 4.1.4)

- 11) Live vaccination
- 12) Any botanical preparation (eg, herbal supplements or traditional Chinese medicines derived from plants, minerals, or animals) intended to treat psoriasis or other immunological diseases.

No concomitant medications (prescription, over-the-counter or herbal) are to be administered during the study unless prescribed for treatment of specific clinical events. Any concomitant therapies must be recorded on the CRF.

The investigator should contact and confirm agreement with the Medical Monitor prior to the administration of any concomitant medications.

#### 6.7.2 Permitted Concomitant Medications

Stable doses of concomitant medication for chronic medical conditions are permitted as long as neither the medication nor the medical condition meet exclusion criteria as detailed in Section 5.2. Dose adjustments of these medications should be avoided during the study unless clinically indicated. If a dose adjustment of these medications should occur, they must be recorded on the Concomitant medications eCRF or the Procedures and Significant non-drug therapies eCRF. The investigator should instruct the subject to notify the study site about any new treatments he/she takes after the start of the study treatment. All medications and significant non-drug therapies (including physical therapy and blood transfusions) administered after the subject starts study treatment must be listed on the Concomitant medications eCRF or the Procedures and Significant non-drug therapies eCRF.

Note: Low potency topical steroids (WHO Class VI and VII) are permitted on the palms, soles, face, and intertriginous areas but should not be used within 24 hours prior to any study visit. Bland emollients (defined as emollients without urea or alpha- or beta-hydroxy acids or other ingredients which are pharmacologically active) are allowed on all body regions but should not be used within 24 hours prior to any study visit.

#### 6.7.3 Rescue Medications

At Week 24, a subject who has may be treated with restricted topicals or shampoos, respectively, as described in Section 6.7.1 at the investigator's discretion. These treatments may be initiated only at Week 24 and not at subsequent time points. A subject who is started on these treatments at Week 24 may use them as needed per the investigator's judgement through Week 52.

### 6.8 Treatment After the End of the Study

At the end of the study, the investigator should ensure that subjects continue to receive appropriate standard of care to treat the condition under study.

In addition, for subjects who continue to demonstrate clinical benefit, BMS may continue to provide study treatment via a rollover extension study requiring approval by responsible health authority and ethics committee, or through another mechanism at the discretion of BMS.

BMS reserves the right to terminate access to BMS supplied study treatment if any of the following occur: a) the study is terminated due to safety concerns; b) the development of BMS-986165 is terminated for other reasons, including but not limited to lack of efficacy and/or not meeting the study objectives; c) the subject can obtain medication from a government sponsored or private health program. In all cases BMS will follow local regulations.

### 7 DISCONTINUATION CRITERIA

### 7.1 Discontinuation from Study Treatment

Subjects MUST discontinue IP (and non-IP at the discretion of the investigator) for any of the following reasons:

- Subject requests to stop study treatment. Subjects who request to discontinue study treatment will remain in the study and must continue to be followed for protocol-specified follow-up procedures. The only exception to this is when a subject specifically withdraws consent for any further contact with him/her or persons previously authorized by subject to provide this information.
- Any clinically significant AE, laboratory abnormality, or intercurrent illness which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject. If treatment is discontinued due to an AE, the AE eCRF must be completed to show that the AE caused discontinuation
- eGFR <45 mL/min on repeat assessment within 7 days
- Abnormal liver tests suggestive of drug-induced liver injury (DILI), as defined in Section 8.2.8 or if the investigator believes that it is in the best interest of the subject
- Subject reports suicidal ideation, suicidal behavior, or suicide attempts at any time after randomization, or documents suicidal ideation by answering "Yes" to Question 4 or 5 on the eC-SSRS, or documents suicidal behavior on the eC-SSRS at any time during the study. The subject should then be immediately referred to a mental health professional for evaluation of suicide risk.

Clinical Protocol BMS-986165

• The subject develops a malignancy with the exception of a subject who develops nonmelanoma skin cancer who may continue in the study at the discretion of the investigator.

- Pregnancy, positive pregnancy test or subject expresses an interest in becoming pregnant (refer to Section 8.2.6)
- Subject develops active TB during the study or prematurely discontinues treatment for LTBI, or subject is noncompliant with LTBI therapy (refer to Section 8.4.4)
- Termination of the study or program by BMS
- Unblinding of a subject's treatment assignment for any reason (emergency or nonemergency)
- Inability or failure to comply with protocol requirements in the opinion of the investigator
- Loss of ability to freely provide consent through imprisonment or involuntary incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness

Refer to the Schedule of Activities (Section 1.3) for data to be collected at the time of treatment discontinuation and follow-up and for any further evaluations that can be completed.

All subjects who discontinue BMS-986165 should comply with protocol-specified follow-up procedures as outlined in Section 1.3. The only exception to this requirement is when a subject withdraws consent for all study procedures including posttreatment study follow-up or loses the ability to consent freely (ie, is imprisoned or involuntarily incarcerated for the treatment of either a psychiatric or physical illness). Replacement of subjects is not permitted.

If study treatment is discontinued prior to the subject's completion of the study, the reason for the discontinuation must be documented in the subject's medical records and entered on the appropriate eCRF page.

### 7.1.1 Temporary Discontinuation of Study Medication

Temporary study treatment discontinuation is allowed only if the subject develops an AE which, in the opinion of the investigator, indicates that it is in the subject's best interest that the study treatment be placed on hold. Study treatment in this situation should be stopped until the AE is medically treated and/or has resolved per PI judgement.

Any temporary study treatment discontinuation as well as restart must be documented on the corresponding eCRF.

# 7.1.2 Post-Study Treatment Follow-up

Post-study follow-up is of critical importance and is essential to preserving subject safety and the integrity of the study. Subjects who discontinue study treatment must continue to be followed for collection of outcomes and/or survival follow-up data as required and in line with Section 4 until death or the conclusion of the study.

Subjects who discontinue study treatment should be encouraged to undergo the Week 52/Early Termination visit and the safety follow-up visit (Section 1.3) in order to support the final efficacy and safety analysis.

Revised Protocol No.: 05 Date: 11-Nov-2020 IM011065

TYK2 Inhibitor

# 7.2 Discontinuation from the Study

Subjects who request to discontinue study treatment will remain in the study and must continue to be followed for protocol specified follow-up procedures as specified in Section 1.3. The only exception to this is when a subject specifically withdraws consent for any further contact with him/her or persons previously authorized by subject to provide this information.

- Subjects should notify the investigator of the decision to withdraw consent from future follow-up in writing, whenever possible.
- The withdrawal of consent should be explained in detail in the medical records by the investigator and entered on the appropriate CRF page.
- In the event that vital status (whether the subject is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.
- If the subject withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.

### 7.3 Lost to Follow-up

- All reasonable efforts must be made to locate subjects to determine and report their ongoing status. This includes follow-up with persons authorized by the subject.
- Lost to follow-up is defined by the inability to reach the subject after a minimum of **three** documented phone calls, faxes, or emails as well as lack of response by subject to one registered mail letter. All attempts should be documented in the subject's medical records.
- If it is determined that the subject has died, the site will use permissible local methods to obtain date and cause of death.
- If investigator's use of third-party representative to assist in the follow-up portion of the study has been included in the subject's informed consent, then the investigator may use a Sponsor-retained third-party representative to assist site staff with obtaining subject's contact information or other public vital status data necessary to complete the follow-up portion of the study.
- The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information.
- If after all attempts, the subject remains lost to follow-up, then the last known alive date as determined by the investigator should be reported and documented in the subject's medical records.

#### 8 STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and timing are summarized in the Schedule of Activities (Section 1.3) and described in Section 4.1.
- Protocol waivers or exemptions are not allowed.
- All significant safety concerns must be discussed with the Medical Monitor immediately upon occurrence or awareness to determine if the subject should continue or discontinue treatment.

• Adherence to the study design requirements, including those specified in the Schedule of Activities (Section 1.3), is essential and required for study conduct.

- All screening evaluations must be completed and reviewed to confirm that potential subjects
  meet all eligibility criteria before randomization. Randomization should not occur until at least
  8 days after the screening visit to allow collection of PSSD data during screening in order to
  calculate a baseline PSSD score. The investigator will maintain a screening log to record details
  of all subjects screened and to confirm eligibility or record reasons for screening failure, as
  applicable.
- Procedures conducted as part of the subject's routine clinical management (eg, blood count) and obtained before signing of informed consent may be utilized for screening or baseline purposes provided the procedure meets the protocol-defined criteria and has been performed within the timeframe defined in the Schedule of Activities (Section 1.3).
- For several assessments, appropriate training will be provided to investigators and designated personnel at sites. Only those individuals trained and certified to perform these assessments will be performing these assessments during the study

# 8.1 Efficacy Assessments

Every effort must be made to ensure that the same evaluator(s) complete the assessment for each subject. If the evaluator(s) is unable to complete the evaluation, then a qualified individual with overlapping experience may perform the evaluation. Documentation of who performed the evaluation is to be recorded in source documents. Assessments are to be performed at approximately the same time of day throughout the duration of the study.

Baseline assessments must be performed per protocol. Procedures not specified in the protocol that are part of standard care may be performed if they do not interfere with study procedures; any data arising from such procedures are not to be reported in the eCRF.

# 8.1.1 Investigator-administered Assessments

# 8.1.1.1 Static Physician Global Assessment (sPGA)

The sPGA is 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration.<sup>24</sup> The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). All sPGA assessments should be performed by a trained physician (eg, dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients. Every effort should be made to ensure that the physician or designee who performed the sPGA evaluations for a subject at randomization performs the sPGA for that subject at all subsequent visits (see APPENDIX 5).

# 8.1.1.2 Psoriasis Area and Severity Index (PASI)

The PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0–4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks).<sup>25</sup> The PASI produces a numeric score that can range from 0 to 72, with

higher PASI scores denoting more severe disease activity. The PASI can also be used to assess response to treatment. The PASI 50 is the proportion of subjects who experience at least a 50% improvement in PASI score as compared with baseline value. The PASI 75, PASI 90, and PASI 100 are defined similarly. BMS will host a training session prior to initiation of the study to demonstrate proper PASI scoring. All PASI assessments should be performed by a trained physician (dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients (see APPENDIX 6).

### 8.1.1.3 Body Surface Area (BSA)

Measurement of psoriasis BSA involvement is estimated using the handprint method with the size of a subject's handprint (including fingers and thumb) representing 1% of BSA involved.  $^{26,27,28}$  The total BSA = 100% with breakdown by body region as follows: head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), trunk including axillae and groin = 30% (30 handprints), lower extremities including buttocks = 40% (40 handprints). BSA assessments should be performed by a dermatologist or appropriately trained investigator who is experienced in the assessment of psoriasis patients.

## 8.1.1.4 Scalp-Specific Physician's Global Assessment (ss-PGA)

For this assessment in subjects with scalp involvement,<sup>29</sup> scalp lesions are evaluated in terms of clinical signs of redness, thickness, and scaliness and scored on the following 5-point ss-PGA scale:

0 =absence of disease, 1 =very mild disease, 2 =mild disease, 3 =moderate disease, 4 =severe disease.

The ss-PGA should be performed by a dermatologist or appropriately trained investigator who is experienced in the assessment of psoriasis patients. An example of the ss-PGA is provided in APPENDIX 7.



# 8.1.1.6 Physician Global Assessment-Fingernails (PGA-F)

In this assessment,<sup>31</sup> the overall condition of the fingernails is rated on a 5-point scale:

0 = clear, 1 = minimal, 2 = mild, 3 = moderate, and 4 = severe

The PGA-F will be performed only in subjects with psoriatic fingernail involvement to assess severity and subsequent improvement. An example is provided in APPENDIX 9. The PGA-F

should be performed by a dermatologist or appropriately training investigator who is experienced in the assessment of psoriasis patients.



### 8.1.1.8 Palmoplantar PGA (pp-PGA)

This measure will be used for subjects with palmoplantar involvement at baseline.<sup>33</sup> The pp-PGA uses a 5-point (0-4) scale:

0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; and 4 = severe (see APPENDIX 11).

The pp-PGA should be performed by a dermatologist or appropriately trained investigator who is experienced in the assessment of psoriasis patients.



# 8.1.2 Subject-reported Assessments

# 8.1.2.1 Psoriasis Symptoms and Signs Diary (PSSD)

The PSSD is an 11-item subject-reported instrument that assesses severity of symptoms and subject-observed signs commonly associated in plaque psoriasis. <sup>35,36</sup> It has been shown to be reliable and valid in measuring symptoms and signs of subjects with moderate-to-severe plaque psoriasis in the clinic and has strong psychometric properties in assessing treatment effects in clinical trials. <sup>37</sup> The PSSD assesses severity of 5 symptoms (itch, pain, stinging, burning, skin

tightness) and 6 subject-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding) using 0–10 numerical ratings. The severity of each item is rated on an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). Two versions of the PSSD were developed, one with a 24-hour recall period (PSSD-24h) and one with a 7-day recall period. The PSSD-24h will be administered daily in this trial to avoid recall bias with a longer recall period (see APPENDIX 13).

### 8.1.2.2 Dermatology Life Quality Index (DLQI)

The DLQI<sup>38</sup> is a subject reported quality of life index which consists of 10 questions concerning symptoms and feelings, daily activities, leisure, work, school, personal relationships, and treatment during the last week. Each question is scored on a scale of 0 to 3 by a tick box: 0 – "not at all", 1 – "a little", 2 – "a lot", or 3 – "very much". The scores are summed, giving a range from 0 (no impairment of life quality) to 30 (maximum impairment) (see APPENDIX 14).





### 8.1.2.8 Psoriatic Arthritis Screening and Evaluation (PASE) Questionnaire

The PASE questionnaire will be administered at screening in subjects with peripheral joint complaints. The PASE questionnaire is a self-administered tool that is used to screen for psoriatic arthritis among subjects who have psoriasis. The PASE questionnaire consists of 15 questions subdivided into 7 questions focusing on symptoms of psoriatic arthritis, and 8 questions focusing on the impact of psoriatic arthritis on function. Each question is scored on a 1-5 scale, with a maximum score of 75. A score of 47 or above has been shown to distinguish between psoriatic arthritis and non-psoriatic arthritis. This questionnaire is only intended to be a screening tool for psoriatic arthritis and does not replace a comprehensive musculoskeletal exam performed by a rheumatologist. The PASE questionnaire should take 6 to 10 minutes to complete and is done only at screening (See APPENDIX 20).

#### 8.2 Adverse Events

The definitions of an AE and SAE can be found in APPENDIX 3.

All AEs will be reported by the subject (or, when appropriate, by a caregiver, surrogate, or the subject's legally authorized representative).

The investigator and any designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study treatment or the study, or that caused the subject to discontinue before completing the study.

Contacts for SAE reporting are specified in APPENDIX 3.

#### 8.2.1 Adverse Events of Interest

Adverse events of interest (AEIs) are AEs for a particular product or class of products that a Sponsor may wish to monitor carefully. Adverse events of interest may be serious or non-serious. Such events may require further investigation to better characterize and understand them. In the BMS-986165 clinical development program, certain skin-related AEs (eg, acne), infection AEs, and CK elevation have been identified as potential AEIs; however, there has been no definitive assessment on the causal relationship between these events and treatment with BMS-986165. Additionally, given a potential association between treatment for autoimmune diseases and increased risk for cancer, malignancy has been identified as a potential AEI. Therefore, additional information about certain skin-related AEs, infection AEs, CK elevation, and malignancy may be collected on the case report form in order to better characterize and understand them.

### 8.2.2 Time Period and Frequency for Collecting AE and SAE Information

The collection of nonserious AE information should begin at initiation of study treatment until discharge from the study (ie, final study visit for a given subject), at the timepoints specified in the Schedule of Activities (Section 1.3).

The Reference Safety Information in Sections 5.6.1 and 5.6.2 of the IB should be used to determine expectedness of SAEs for expedited reporting. Following the subject's written consent to participate in the study, all SAEs, whether related or not related to study drug, must be collected, including those thought to be associated with protocol-specified procedures.

All SAEs must be collected from the date of subject's written consent until 30 days after the final dose of the study drug or subject's participation in the study if the last scheduled visit occurs at a later time. Monitoring for SAEs will occur at every study visit.

- The investigator must report any SAE that occurs after these time periods and that is believed to be related to study drug or protocol-specified procedure. Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded on the appropriate section of the CRF.
- All SAEs will be recorded and reported to Sponsor or designee within 24 hours, as indicated in APPENDIX 3.
- The investigator will submit any updated SAE data to the sponsor within 24 hours of this being available.

Investigators are not obligated to actively seek AEs or SAEs in former study subjects; however, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he/she considers the event reasonably related to the study treatment or study participation, the investigator must promptly notify the Sponsor.

The method of evaluating and assessing causality of AEs and SAEs and the procedures for completing and reporting/transmitting SAE reports are provided in APPENDIX 3.

### 8.2.3 Method of Detecting AEs and SAEs

Adverse events can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a subject. (In order to prevent reporting bias, subjects should not be questioned regarding the specific occurrence of one or more AEs.)

### 8.2.4 Follow-up of AEs and SAEs

- Nonserious AEs should be followed to resolution or stabilization, or reported as SAEs if they become serious (see APPENDIX 3).
- Follow-up is also required for nonserious AEs that cause interruption or discontinuation of study treatment and for those present at the end of study treatment as appropriate.
- All identified nonserious AEs must be recorded and described on the nonserious AE page of the CRF. Completion of supplemental CRFs may be requested for AEs and/or laboratory abnormalities that are reported/identified during the course of the study.
- After the initial AE/SAE report, the investigator is required to proactively follow each subject at subsequent visits/contacts. All SAEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the subject is lost to follow-up (as defined in Section 7.3).

Further information on follow-up procedures is given in APPENDIX 3.

### 8.2.5 Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the Sponsor of SAEs is essential so that legal obligations and ethical responsibilities towards the safety of subjects and the safety of a product under clinical investigation are met.
- An investigator who receives an investigator safety report describing SAEs or other specific safety information (eg, summary or listing of SAEs) from the Sponsor will file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

Sponsor or designee will be reporting AEs to regulatory authorities and ethics committees according to local applicable laws including European Directive 2001/20/EC, FDA Code of Federal Regulations 21 CFR Parts 312 and 320, and Standard and Procedure for Expedited Reporting of Safety Data during Clinical Trials of Drugs, issued by the CDE. A SUSAR (Suspected, Unexpected Serious Adverse Reaction) is a subset of SAEs and will be reported to the appropriate regulatory authorities and investigators following local and global guidelines and requirements.

# 8.2.6 Pregnancy

In the event a subject becomes pregnant during the trial, the study treatment must be discontinued immediately. If the subject becomes pregnant while on treatment or within 3 days of discontinuing study treatment, the investigator must immediately notify Drug Safety of this event and complete and forward a Pregnancy Surveillance Form to Drug Safety within 24 hours of awareness of the event and in accordance with SAE reporting procedures described in APPENDIX

3. The investigator must also notify the Medical Monitor or designee of this event within 24 hours of awareness of pregnancy.

The pregnant subject will need to be followed up until the conclusion of the pregnancy for pregnancy outcomes. The safety data of the subject will continue to be collected under the same rules as instructed in Section 7.1.

Any pregnancy that occurs in a female partner of a male study subject should be reported to Drug Safety. In order for Sponsor or designee to collect any pregnancy surveillance information from the female partner, the female partner must sign an ICF for disclosure of this information. Information on this pregnancy will be collected on the Pregnancy Surveillance Form.

### 8.2.7 Laboratory Test Result Abnormalities

The following laboratory test result abnormalities should be captured on the nonserious AE CRF page or SAE Report Form electronic, as appropriate. Paper forms are only intended as a back-up option when the electronic system is not functioning.

- Any laboratory test result that is clinically significant or meets the definition of an SAE
- Any laboratory test result abnormality that required the subject to have study treatment discontinued or interrupted
- Any laboratory test result abnormality that required the subject to receive specific corrective therapy

It is expected that wherever possible, the clinical rather than laboratory term would be used by the reporting investigator (eg, anemia versus low hemoglobin value).

# 8.2.8 Potential Drug Induced Liver Injury (DILI)

All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs (see Section 8.2 and APPENDIX 3 for reporting details). Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential DILI event.

Potential DILI is defined as:

1) ALT or AST elevation >3 times ULN

#### **AND**

2) Total bilirubin >2 times ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase),

#### **AND**

3) No other immediately apparent possible causes of liver function test elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic.

# 8.2.9 Other Safety Considerations

Any significant worsening of a pre-existing medical condition noted during interim or final physical examinations, electrocardiogram, x-ray filming, any other potential safety assessment required or not required by protocol should also be recorded as a nonserious or serious AE, as appropriate, and reported accordingly.

#### 8.3 Overdose

For this study, taking more than 2 days' worth of study medication within a 24-hour time period will be considered an overdose.

In the event of an overdose the investigator should:

- 1) Contact the Medical Monitor immediately
- 2) Closely monitor the subject for AEs/SAEs and laboratory abnormalities

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the Medical Monitor based on the clinical evaluation of the subject.

### 8.4 Safety

Planned time points for all safety assessments are listed in the Schedule of Activities (Section 1.3).

### 8.4.1 Physical Examinations

A complete physical examination will include general appearance, vital signs, eyes, ears, nose mouth, throat, neck, respiratory, cardiovascular, respiratory, GI, lymphatic, musculoskeletal, skin, psychiatric and neurologic exams. A targeted physical examination will include vital signs, and any organ system associated with an AE or a laboratory abnormality.

### 8.4.2 Vital Signs

Refer to Schedule of Activities (Section 1.3).

### 8.4.3 Electrocardiograms

A 12-lead ECG will be performed at the visits indicated in the Schedule of Activities (Section 1.3). The patient will remain supine for 5-10 minutes prior to the ECG and must have their lab work done after the tracing so that the ECG results remain as accurate as possible. The ECG results will be read by the primary study investigator or a designee.

### 8.4.4 Tuberculosis Screening and Chest Imaging

Chest imaging results and PE are part of the process to assess a subject's eligibility, as outlined in Section 1.3 and as defined in exclusion criterion 3.c (Section 5.2). Chest imaging (eg, chest x-ray, chest CT scan) at the screening visit is required if not already performed and documented within 6 months of obtaining written informed consent. A subject must not have active signs or symptoms of TB, as judged by the investigator, to be eligible for the study.

In addition to a complete PE and medical history to evaluate exposure to TB, all subjects will have a screening test, an IGRA (eg, QuantiFERON®-TB test) performed centrally. If unable to obtain

central laboratory results, an IGRA test could be obtained locally, after consultation with the Medical Monitor. A subject with an indeterminate IGRA test result must be retested for confirmation. If the second result is again indeterminate, the subject will be excluded from the study. If the second result is positive, the subject should be treated as having LTBI provided there are no signs or symptoms of active TB. If the second result is negative, the subject may be eligible provided no other exclusion criterion for TB is met.

### 8.4.5 Clinical Safety Laboratory Assessments

Investigators must document their review of each laboratory safety report

| Hematology | |
|---|---|
| Hemoglobin (Hgb) | |
| Hematocrit (Hct) | |
| White Blood Cell Count, including differential | |
| Platelet Count | |
| Chemistry | |
| A C/T | T (1D () |
| AST | Total Protein |
| ALT | Albumin |
| Total Bilirubin | Sodium |
| Direct Bilirubin (if total bilirubin >ULN) | Potassium |
| Alkaline Phosphatase | Chloride |
| Lactate Dehydrogenase (LDH) | Calcium |
| Creatinine | Phosphorus |
| Blood Urea Nitrogen (BUN) | Creatine Kinase (CPK)* |
| Uric Acid | Estimated Glomerular Filtration Rate (eGFR) |
| Glucose (fasting at some visits) | |

### Urinalysis

Protein

Glucose

Blood

Leukocyte Esterase

Specific Gravity

pН

Microscopic Examination (reflex if abnormal)

# **Lipid Panel**

Cholesterol (total)

High Density Lipoprotein (HDL)

Low Density Lipoprotein (LDL)

**Triglycerides** 

### **Infectious Serologies**

(HIV RNA as appropriate)

Hepatitis C Antibody with reflex to Hepatitis C RNA if positive

Hepatitis B Surface Antigen (HBsAg)

Hepatitis B Surface Antibody (HBsAb)

Hepatitis B Core Antibody (HBcAb)

Hepatitis B DNA Viral Load (HBV-DNA)

HIV-1 and -2 antibody

# **Other Analyses**

Pregnancy test (WOCBP only: serum hCG test at screening, followed by urine hCG test or serum hCG test every 4 weeks)

Follicle Stimulating Hormone (FSH) (to confirm menopausal status [see APPENDIX 4], at screening) use as applicable

Hemoglobin A1C

Thyroid Stimulating Hormone (TSH)

• If TSH above normal reference range, test free T4; if TSH below normal range, test free T4 & T3

High Sensitivity C Reactive Protein (hsCRP)

Serum immunoglobulin (IgM, IgG, IgA, IgE)

\*If CK >2.5 × ULN, then reflex testing (ie, CK-MB, Troponin I) will be required.

### 8.4.5.1 Estimated Glomerular Filtration Rate (eGFR)

Glomerular filtration rate will be estimated using the Modification of Diet in Renal Disease (MDRD) equation at screening and during the study at selected visits.

The MDRD equation is as follows:<sup>45</sup>

eGFR = 
$$175 \times \text{standardized SCr}^{-1.154} \times \text{age}^{-0.203} \times 1.212$$
 [if black] or 0.742 [if female]

Note: GFR is expressed as mL/min/1.73 m<sup>2</sup> of body surface area and SCr (serum creatinine) is expressed in mg/dL.

Subjects with an eGFR <45 mL/min will be excluded from participation

# 8.4.6 Depression Monitoring

Depression will be monitored by administration of the eight-item Patient Health Questionnaire (PHQ-8) at screening and during visits as outlined in Section 1.3.

# 8.4.6.1 Eight Item Patient Health Questionnaire (PHQ-8)

The PHQ-8 is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies. <sup>46</sup> Each of the 8 questions is based on a 2-week recall and scored on a scale of 0 to 3 by a tick box as: Not at All, Several Days, More than Half the Days and Nearly Every Day. A score of  $\geq$ 10 is suggestive of moderate depressive symptoms (see APPENDIX 21). <sup>47</sup> If a subject scores  $\geq$  15 on the PHQ-8 during the study, the investigator will review the situation and refer the subject to a mental health professional if deemed necessary.

### 8.4.7 Suicidal Ideation and Behavior (SIB) Monitoring

Subjects in this clinical trial will be monitored for SIB by the eC-SSRS (Section 8.4.7.1) at the visits outlined in the Schedule of Activities (Section 1.3). Subjects who answer yes to Questions 4 or 5 which indicates a suicidal ideation severity level of 4 or 5 or document suicidal behavior or suicidal attempts on the eC-SSRS will have their treatments discontinued and be immediately referred to a mental health professional for further evaluation. In addition, family members or caregivers of the subjects will be instructed to immediately report any suicidal ideation, suicidal behavior, or suicide attempt to the investigator.

### 8.4.7.1 Electronic Columbia Suicide Severity Rating Scale (eC-SSRS)

The electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) is a computer-automated, patient-reported version of the C-SSRS instrument that defines 11 categories of SIB events. 48,49,50 The categories are as follows:

- Suicidal ideation
  - 1) Passive
  - 2) Active: Nonspecific (no method, intent, or plan)
  - 3) Active: Method, but no intent or plan
  - 4) Active: Method and intent, but no plan
  - 5) Active: Method, intent, and plan
- Suicidal behavior
  - 1) Completed suicide
  - 2) Suicide attempt
  - 3) Interrupted attempt
  - 4) Aborted attempt
  - 5) Preparatory actions toward imminent suicidal behaviors
  - Self-injurious behavior, no suicidal intent

Definitions of these categories can be found in APPENDIX 22<sup>51</sup>







# 8.6 Health Economics OR Medical Resource Utilization and Health Economics

Health Economics/Medical Resource Utilization and Health Economics parameters will not be evaluated in this study.

#### 9 STATISTICAL CONSIDERATIONS



### 9.2 Populations for Analyses

For purposes of analysis, the following analysis sets will be used in this study:

Enrolled Population: All subjects who sign informed consent.

**Full Analysis Set (FAS):** All subjects who were randomized. Following the intent-to-treat principle, subjects will be analyzed according to the treatment group assigned at randomization. The FAS will be the primary efficacy analysis population.

**Per Protocol Set (PPS):** A subset of the FAS who are compliant with study treatment and who do not have any relevant protocol deviations that may impact the coprimary efficacy endpoint assessments (Section 9.6.3). The PPS will be analyzed for the coprimary endpoint comparisons according to the treatment assigned at randomization.

**As-treated Population:** All randomized subjects who took at least one dose of study treatment. Subjects will be analyzed according to treatment received. The As-treated population will be for safety analyses.

### 9.3 Endpoints

### 9.3.1 Primary Endpoints

The coprimary efficacy endpoints for BMS-986165 compared to placebo at Week 16 are defined as:

- sPGA 0/1 response assessed as a proportion of subjects with a sPGA score of 0 or 1
- PASI 75 response assessed as a proportion of subjects who achieve a 75% improvement from baseline in the PASI score

# 9.3.2 Key Secondary Endpoints

The key secondary endpoints for BMS-986165 compared to placebo at Week 16 are defined as:

- PASI 90 response assessed as a proportion of subjects who achieve a 90% improvement from baseline in the PASI score
- sPGA 0 response assessed as a proportion of subjects with a sPGA score of 0
- PASI 100 response assessed as a proportion of subjects who achieve a 100% improvement from baseline in the PASI score
- Change from baseline in PSSD symptom score
- PSSD symptom score of 0 assessed as a proportion of subjects with a PSSD symptom score of 0 among subjects with a baseline PSSD symptom score ≥1
- ss-PGA 0/1 assessed as a proportion of subjects with a ss-PGA score 0 or 1 among subjects with a baseline ss-PGA score >3
- DLQI 0/1 assessed as a proportion of subjects with a DLQI score of 0 or 1 among subjects with a baseline DLQI score >2
- PGA-F 0/1 assessed as a proportion of subjects with a PGA-F score of 0 or 1 among subjects with a baseline PGA-F score >3
- pp-PGA 0/1 assessed as a proportion of subjects with a pp-PGA score of 0 or 1 among subjects with a baseline pp-PGA score ≥3





Clinical Protocol BMS-986165

### 9.4 Efficacy Analyses

Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified. Efficacy values will be summarized for all visits in which the variable is assessed. Details of the planned analyses of endpoints during the 16-week double-blind placebo-controlled period will be documented in the statistical analysis plan (SAP) and finalized before the Week 16 database lock.

During the first 16 weeks of treatment, data will be presented for the following treatments:

- BMS-986165 6 mg QD
- Placebo

After Week 16, data will be presented for the following treatments:

- BMS-986165 6 mg QD
- Placebo —BMS-986165 6 mg QD (starting from Week 16 through Week 52)
- All BMS-986165 6 mg QD (all subjects exposed to BMS-986165 6 mg QD; includes subjects on placebo that switched to BMS-986165 6 mg QD)

### 9.4.1 Coprimary Endpoint Analyses

The analysis model for the coprimary efficacy endpoints, sPGA 0/1 and PASI 75 (responder/nonresponder) at Week 16, will use stratified Cochran-Mantel-Haenszel (CMH) tests stratified by the stratification factors used for randomization (see Section 4.1.2) to compare the response rates of BMS-986165 6 mg QD to placebo using the Week 16 data of the FAS. The odds ratio (ratio of odds in BMS-986165 6 mg QD group to the odds in placebo group) and the corresponding 2-sided 95% confidence interval (CI) will be provided. Estimates of proportions and their 2-sided 95% CIs will be provided.

### 9.4.1.1 Imputation Methods for Coprimary Endpoints

Non-responder imputation (NRI) will be used for coprimary efficacy endpoints for subjects who discontinue treatment or study prior to Week 16, start a protocol prohibited medication/therapy that could improve psoriasis during the first 16 weeks of treatment, or who have otherwise missing endpoint data at the specified timepoint. NRI will be the primary method of imputation for the coprimary efficacy endpoints.

# 9.4.1.2 Sensitivity Analyses for the Coprimary Endpoints

Sensitivity analyses to be performed for the coprimary endpoints will be described in the SAP prior to the Week 16 database lock.

### 9.4.1.3 Supportive Analyses for the Coprimary Endpoints

The coprimary efficacy endpoints will be analyzed using the Week 16 data of the PPS using the analysis described in Section 9.4.1 and the imputation methods described in Section 9.4.1.1.

Additionally, the coprimary efficacy endpoints for the FAS will be analyzed with a logistic regression model with treatment and the stratification factors used for randomization as covariates.

### 9.4.1.4 Subgroup Analyses for the Coprimary Endpoints

Subgroup analyses will be conducted for the coprimary efficacy endpoints for the FAS using the analysis described in Section 9.4.1 and the imputation methods described in Section 9.4.1.1. Subgroups to be evaluated may include the following:

- Gender
- Age categories (<65;  $\ge65$ )
- Prior biologic use (yes/no)
- Prior systemic treatment of psoriasis (yes/no)
- Country

Additional subgroups may be defined for descriptive summaries in the SAP.

### 9.4.2 Secondary Endpoint Analyses

The analysis model for the binary secondary endpoints will use stratified CMH tests stratified by the stratification factors used for randomization (see Section 4.1.2) to compare the response rates of BMS-986165 6 mg QD to placebo for the FAS. The odds ratio (ratio of odds in BMS-986165 6 mg QD group to the odds in placebo group) and the corresponding 2-sided 95% CI will be provided.

The analysis model for continuous secondary endpoints will use analysis of covariance (ANCOVA) with treatment and stratification factors used for randomization as fixed effects. The baseline value will be added into the model as a covariate. Treatment differences based on least-squares (LS) means and the corresponding 2-sided 95% CIs will be provided for the difference between BMS-986165 6 mg QD and placebo.

# 9.4.2.1 Imputation Methods for Secondary Endpoints

The NRI will be applied to the analyses of binary secondary efficacy endpoints for subjects who discontinue early, start a protocol prohibited medication/therapy that could improve psoriasis, or who have otherwise missing endpoint data prior to the specified timepoint.

For continuous secondary efficacy endpoints, a modified baseline observation carried forward (mBOCF) will be used for missing data. The baseline observation will be carried forward for subjects who discontinue study treatment due to:

- Lack of efficacy
- AEs

and for subjects who start a protocol prohibited medication/therapy that could improve psoriasis prior to the endpoint. The last valid observation will be carried forward for all other subjects with missing data.



### 9.5 Safety Analyses

Safety data will be analyzed for AEs, SAEs, laboratory analytes, vital signs, ECGs, and suicidality and depression. Safety will be summarized using the As-treated population. Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified.

During the first 16 weeks of treatment data will be presented for the following treatments:

- BMS-986165 6 mg QD
- Placebo

After Week 16 data will be presented for the following treatments:

- BMS-986165 6 mg QD
- Placebo→BMS-986165 6 mg QD (starting from Week 16 through Week 52)
- All BMS-986165 6 mg QD (all subjects exposed to BMS-986165 6 mg QD; includes subjects on placebo that switched to BMS-986165 6 mg QD)

#### 9.5.1 Adverse Events

Treatment-emergent adverse events (TEAEs), SAEs and deaths, and AEs leading to study treatment discontinuation, AEs by maximum severity, and AEs by relationship will be summarized by the MedDRA system organ class and preferred term. All TEAEs, AEIs, as well each AE adjudicated category (ie, infections, cardiovascular, and suicidal ideation and behavior) will also be summarized by preferred term sorted by decreasing frequency.

### 9.5.2 Vital Signs and ECGs

Vital signs and ECGs will be summarized as raw, change from baseline, and change from maximum postbaseline value. Incidence of abnormal ECG will also be summarized.

### 9.5.3 Clinical Laboratory Tests

Laboratory analytes will be summarized as raw, change from baseline, and change from maximum postbaseline value. Incidence of abnormal, high, or low values will be summarized.

### 9.5.4 Suicidality and Depression Assessments

Suicidality and depression will be assessed using eC-SSRS and PHQ-8. Data will be summarized, as applicable.

### 9.6 Other Analyses

### 9.6.1 Demographics and Baseline Data

Demographics and baseline data will be summarized by treatment for each applicable analysis population. Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified.

#### 9.6.2 Prior and Concomitant Medications

Prior and concomitant medications, categorized by medication group and subgroup according to the World Health Organization (WHO) Drug Dictionary, will be summarized by treatment for the As-treated population. Medications with an end date prior to the first dose of study drug will be considered prior medications.

#### 9.6.3 Relevant Protocol Deviations

Relevant protocol deviations are deviations that can have an impact on the primary efficacy endpoints. The impact of relevant protocol deviations on the primary efficacy results will be assessed by excluding subjects from the FAS to define the PPS in supportive analyses of the primary efficacy endpoints. Relevant protocol deviations to be considered regarding exclusion of subjects from the FAS will include the following:

- Subject was randomized but did not take any study treatment
- Subject failed to meet any study inclusion criteria but was randomized to receive study treatment
- Subject met a study exclusion criterion which may have an impact on the coprimary efficacy endpoints but was randomized to receive study treatment
- Subject was noncompliant with study treatment within the first 16 weeks of treatment; defined as <80% compliant with study treatment
- Subject took prohibited concomitant medication prior to Week 16
- Subject received treatment different than assigned treatment at any visit prior to Week 16

All subjects with relevant protocol deviations will be identified prior to the Week 16 database lock. Relevant protocol deviations will be summarized by treatment group and deviation category for the FAS population.

# 9.7 Interim Analyses

No interim analysis is currently planned.

# 9.8 Analysis and Reporting

An unblinded analysis of the data collected up to Week 16 will be conducted once all randomized subjects have either completed the placebo-controlled treatment period (ie, through Week 16) or have discontinued prior to Week 16. Details of these analyses will be provided in an SAP that will be finalized before the Week 16 database lock. A final database lock and analysis will occur after all subjects complete Week 52 or discontinue prior to Week 52.

#### 10 REFERENCES

Parisi R, Symmons DP, Griffiths CE, et al. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol 2013;133(2):377-85.

- <sup>2</sup> Kupetsky EA, Keller M. Psoriasis vulgaris: an evidence-based guide for primary care. J Am Board Fam Med 2013;26(6):787-801.
- World Health Organization. Global Report on psoriasis. WHO 2016.
- <sup>4</sup> Langley RG, Krueger GG, Griffiths CE. Psoriasis: epidemiology, clinical features, and quality of life. Ann Rheum Dis 2005;64:18-25.
- Oueiro R, Tejón P, Alonso S, Coto P. Age at disease onset: a key factor for understanding psoriatic disease. Rheumatology (Oxford) 2014;53(7):1178-85.
- Mrowietz U, Kragballe K, Reich K, et al. Definition of treatment goals for moderate to severe psoriasis: a European consensus. Arch Dermatol Res. 2011 Jan;303(1):1-10.
- Nestle FO, Kaplan DH, Barker J. Mechanisms of Disease: Psoriasis. N Engl J Med 2009;361:496-509.
- <sup>8</sup> Langley RG, Kreuger GG, Griffiths CE. Psoriasis: epidemiology, clinical features, and quality of life. Ann Rheum Dis 2005;64(Suppl II):ii18–ii23.
- Mehta NN, Afzar RS, Shin DB, Neimann AL, Troxel AB, Gelfand JM. Patients with severe psoriasis are at increased risk of cardiovascular mortality: cohort study using the General Practice Research Database. European Heart J 2010;31:1000–1006.
- Novartis. Rheumatrex® (methotrexate). United States Prescribing Information. 2016.
- Novartis. Neoral® (cyclosporine). United States Prescribing Information. 2009.
- <sup>12</sup> Celgene. Otezla® (apremilast). United States Prescribing Information. 2017.
- Abbvie. Humira® (adalimumab). United States Prescribing Information. 2017.
- <sup>14</sup> Janssen Biotech. Remicade® (infliximab). United States Prescribing Information. 2013.
- <sup>15</sup> Janssen Biotech. Stelara® (ustekinumab). United States Prescribing Information. 2016.
- <sup>16</sup> Novartis. Cosentyx<sup>®</sup> (sekukinumab). United States Prescribing Information. 2015.
- <sup>17</sup> Eli Lilly. Taltz<sup>®</sup> (ixekizumab). United States Prescribing Information. 2017.
- <sup>18</sup> Valeant. Siliq® (brodalumab). United States Prescribing Information. 2017.
Armstrong AW, Robertson AD, Wu J, Schupp C, Lebwohl MG. Undertreatment, Treatment Trends, and Treatment Dissatisfaction Among Subjects with Psoriasis and Psoriatic Arthritis in the United States. Findings from the National Psoriasis Foundation Surveys, 2003-2011. JAMA Dermatol 2013;149(10):1180–1185.

- Watford WT, Hissong BD, Bream JH, et al. Signaling by IL-12 and IL-23 and the immunoregulatory roles of STAT4. Immunol Rev. 2004;202:139-56.
- Tokarski JS, Zupa-Fernandez A, Tredup JA, et al.. Tyrosine Kinase 2-Mediated Signal Transduction in T Lymphocytes Is Blocked by Pharmacological Stabilization of its Pseudokinase Domain. J Biol Chem 2015;290:11061-11074.
- Shaw MH, Boyartchuk V, Wong S, et al. A natural mutation in the Tyk2 pseudokinase domain underlies altered susceptibility of B10.Q/J mice to infection and autoimmunity. Proc Natl Acad Sci U S A. 2003;100:11594-11599.



- <sup>24</sup> Feldman SR, Krueger GG. Psoriasis assessment tools in clinical trials. Ann Rheum Dis 2005;64:ii65-ii68.
- Fredriksson T, Pettersson U. Severe psoriasis-oral therapy with a new retinoid. Dermatologica 1978;157(4):238-44.
- <sup>26</sup> Rossiter ND, Chapman P, Haywood IA. How big is a hand? Burns. 1996;22:230-1.
- Thomas CL, Finlay AY. The 'handprint' approximates to 1% of the total body surface area whereas the 'palm minus the fingers' does not. Br J Dermatol. 2007;157(5):1080-1.
- Long CC, Finlay AY, Averill RW. The rule of hand: 4 hand areas = 2 FTU = 1 g. Arch Dermatol. 1992;128:1129–30.
- Kragballe K, Menter A, Lebwohl M, et al. Long-term management of scalp psoriasis: perspectives from the international psoriasis council. J Dermatol Treat. 2013;24:188-192.



- Tan EST, Chong W-S, Liang Tey H. Nail psoriasis: a review. Am J Clin Dermatol. 2012;13:375-388.
- Bissonnette R, Pariser DM, Wasel NR, et al. Apremilast, an oral phosphodiesterase-4 inhibitor, in the treatment of palmoplantar psoriasis: Results of a pooled analysis from phase II PSOR-005 and phase III Efficacy and Safety Trial Evaluating the Effects of Apremilast in Psoriasis

(ESTEEM) clinical trials in patients with moderate to severe psoriasis. J Am Acad Dermatol. 2016;75:99-105.

- Feldman SR. Development of a patient-reported outcome questionnaire for use in adults with moderate-to-severe plaque psoriasis: The Psoriasis Symptoms and Signs Diary. Journal of Dermatology & Dermatologic Surgery. 2016;20:19–26.
- Mathias SD. Measurement properties of a patient-reported outcome measure assessing psoriasis severity: The psoriasis symptoms and signs diary. Journal of Dermatological Treatment. 2016;27(4):322-327.
- Armstrong A, Puig L, Langley R, et al. Validation of psychometric properties and development of response criteria for the Psoriasis Symptoms and Signs Diary (PSSD): results from a phase III clinical trial. Journal of Dermatological Treatment. 2017: 1-31. DOI: 10.1080/09546634.2017.1364694.
- Finlay, AY, Khan, GK: Dermatology Life Quality Index (DLQI): A simple practical measure for routine clinical use. Clin Exp Dermatol. 1994;19:210–216.
- Husni ME, Meyer KH, Cohen DS, Mody E, Qureshi AA. J Am Acad Dermatol 2007;57(4):581-7
- Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, et al. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med 2006;145(4):247–54.
- Kroenke K, Strine TW, Spitzer RL, et al. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009;114(1-3):163-173.
- Dhingra SS, Kroenke K, Zack MM, Strine TW, Balluz LS. PHQ-8 Days: a measurement option for DSM-5 Major Depressive Disorder (MDD) severity. Population Health Metrics. 2011;9:11. doi:10.1186/1478-7954-9-11.

Clinical Protocol BMS-986165

The Federal Register. Guidance for Industry- Suicidal ideation and behavior: prospective assessment of occurrence in clinical trials. (06-Aug-2012). https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM225130.pdf. Accessed 22-Mar-2018.

- <sup>49</sup> Greist JH, Mundt JC, Gwaltney CJ, Jefferson JW, Posner K. Predictive value of baseline electronic Columbia–Suicide Severity Rating Scale (eC–SSRS) assessments for identifying risk of prospective reports of suicidal behavior during research participation. Innov Clin Neurosci. 2014;11(9–10):23–31.
- Mundt JC, Greist JH, Jefferson JW, Federico M, Mann JJ, Posner K. Prediction of suicidal behavior in clinical research by lifetime suicidal ideation and behavior ascertained by the electronic Columbia-Suicide Severity Rating Scale. J Clin Psychiatry. 2013;74(9):887-893.
- Posner, K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): Classification of Suicidal Events in the FDA's Pediatric Suicidal Risk Analysis of Antidepressants. Am J Psychiatry. 2007;164:1035-1043
- <sup>52</sup> Collins SL, Moore RA, McQuay HJ. The visual analogue pain intensity scale: what is moderate pain in millimetres? Pain. 1997;72(1-2):95-7.

Revised Protocol No.: 05 Date: 11-Nov-2020 IM011065

TYK2 Inhibitor

75

# 11 APPENDICES

# APPENDIX 1 ABBREVIATIONS AND TRADEMARKS

| Term | Definition |
|----------|--------------------------------------|
| AE | adverse event |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| ANOVA | analysis of variance |
| Anti-HCV | hepatitis C virus antibody |
| AST | aspartate aminotransferase |
| BID | twice daily |
| BMS | Bristol-Myers Squibb |
| BOCF | baseline observation carried forward |
| BSA | body surface area |
| BUN | blood urea nitrogen |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CMH | Cochran-Mantel-Haenszel |
| CK | creatine kinase |
| DILI | drug-induced liver injury |
| DLQI | Dermatology Life Quality Index |
| DMC | Data Monitoring Committee |
| ECG | electrocardiogram |

| Term | Definition |
|---------|------------------------------------------------------|
| eCRF | electronic case report form |
| eC-SSRS | electronic Columbia-Suicide Severity Rating<br>Scale |
| eGFR | Estimated Glomerular Filtration Rate |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| FSH | follicle-stimulating hormone |
| HBcAb | hepatitis B core antibody |
| HBsAb | hepatitis B surface antibody |
| HBsAg | hepatitis B surface antigen |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| Hgb | hemoglobin |
| HIV | human immunodeficiency virus |
| hs-CRP | high-sensitivity C-reactive protein |
| IB | Investigator Brochure |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IFN | interferon |
| ΙΓΝγ | interferon gamma |
| IgG | immunoglobulin gamma |
| IGRA | interferon gamma release assay |
| IL | interleukin |
| IMP | investigational medicinal product |
| IP | investigational product |
| IRT | interactive response technology |

| Term | Definition |
|--------|-----------------------------------------------|
| ITT | intent-to-treat |
| IV | intravenous |
| JAK | Janus kinase |
| LOCF | last observation carried forward |
| LS | least-squares |
| LTBI | latent tuberculosis infection |
| MACE | Major Adverse Cardiovascular Event |
| mBOCF | modified baseline observation carried forward |
| NRI | non-responder imputation |
| NSAID | nonsteroidal anti-inflammatory drug |
| PASE | psoriatic arthritis screening and evaluation |
| PASI | Psoriasis Area and Severity Index |
| PD | pharmacodynamics |
| PE | physical examination |
| PGA-F | Physician Global Assessment-Fingernails |
| PHQ-8 | Eight Item Patient Health Questionnaire |
| PK | pharmacokinetics |
| pp-PGA | palmoplantar Physician's Global Assessment |
| PPS | Per Protocol Set |
| PRO | patient reported outcome |
| PsA | psoriatic arthritis |
| PSSD | Psoriasis Symptoms and Signs Diary |
| QD | once daily |
| QOD | every other day |
| RBC | red blood cell |
| RNA | ribonucleic acid |

| Term | Definition |
|--------|--------------------------------------------------|
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SIB | Suicidal Ideation and Behavior |
| SLE | systemic lupus erythematosus |
| sPGA | static Physician Global Assessment |
| ss-PGA | scalp-specific Physician's Global Assessment |
| STAT | signal transducer and activator of transcription |
| ТВ | tuberculosis |
| T4 | thyroxine |
| Т3 | triiodothyronine |
| TEAE | treatment-emergent adverse event |
| TNF | tumor necrosis factor |
| TYK2 | tyrosine kinase 2 |
| ULN | upper limit of normal |
| WOCBP | women of childbearing potential |

Revised Protocol No.: 05

# APPENDIX 2 STUDY GOVERNANCE CONSIDERATIONS REGULATORY AND ETHICAL CONSIDERATIONS GOOD CLINICAL PRACTICE

This study will be conducted in accordance with:

- Good Clinical Practice (GCP),
- as defined by the International Council on Harmonisation (ICH)
- in accordance with the ethical principles underlying European Union Directive 2001/20/EC
- United States Code of Federal Regulations, Title 21, Part 50 (21CFR50)
- applicable local requirements.

The study will be conducted in compliance with the protocol. The protocol and any amendments and the subject informed consent will receive approval/favorable opinion by Institutional Review Board/Independent Ethics Committee (IRB/IEC), and regulatory authorities according to applicable local regulations prior to initiation of the study.

All potential serious breaches must be reported to Sponsor or designee immediately. A serious breach is a breach of the conditions and principles of GCP in connection with the study or the protocol, which is likely to affect, to a significant degree, the safety or physical or mental integrity of the subjects of the study or the scientific value of the study.

Personnel involved in conducting this study will be qualified by education, training, and experience to perform their respective tasks.

This study will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure, debarment).

#### INSTITUTIONAL REVIEW BOARD/INDEPENDENT ETHICS COMMITTEE

Before study initiation, the investigator must have written and dated approval/favorable opinion from the IRB/IEC for the protocol, consent form, subject recruitment materials (eg, advertisements), and any other written information to be provided to subjects. The investigator or BMS should also provide the IRB/IEC with a copy of the Investigator Brochure or product labeling information to be provided to subjects and any updates.

The investigator, Sponsor or designee should provide the IRB/IEC with reports, updates and other information (eg, expedited safety reports, amendments, and administrative letters) according to regulatory requirements or institution procedures.

# COMPLIANCE WITH THE PROTOCOL AND PROTOCOL REVISIONS

The investigator should not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion of an amendment from the IRB/IEC (and if applicable, also by local health authority) except where necessary to eliminate an immediate hazard(s) to study subjects.

If a deviation or change to a protocol is implemented to eliminate an immediate hazard(s) prior to obtaining relevant approval/favorable opinion(s) the deviation or change will be submitted, as soon as possible to:

- IRB/IEC for
- Regulatory Authority(ies), if applicable by local regulations (per national requirements)

Documentation of approval/favorable opinion signed by the chairperson or designee of the IRB(s)/IEC(s) and if applicable, also by local health authority must be sent to BMS.

If an amendment substantially alters the study design or increases the potential risk to the subject: (1) the consent form must be revised and submitted to the IRB(s)/IEC(s) for review and approval/favorable opinion; (2) the revised form must be used to obtain consent from subjects currently enrolled in the study if they are affected by the amendment; and (3) the new form must be used to obtain consent from new subjects prior to enrollment.

If the revision is done via an administrative letter, investigators must inform their IRB(s)/IEC(s).

#### FINANCIAL DISCLOSURE

Investigators and sub-Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### INFORMED CONSENT PROCESS

Investigators must ensure that subjects are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which they volunteer to participate.

In situations where consent cannot be given to subjects, their legally acceptable representatives (as per country guidelines) are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which the subject volunteers to participate.

Sponsor or designee will provide the investigator with an appropriate (ie, Global or Local) sample informed consent form which will include all elements required by ICH, GCP and applicable regulatory requirements. The sample informed consent form will adhere to the ethical principles that have their origin in the Declaration of Helsinki.

Investigators must:

• Provide a copy of the consent form and written information about the study in the language in which the subject is most proficient prior to clinical study participation. The language must be non-technical and easily understood.

- Allow time necessary for subject or subject's legally acceptable representative to inquire about the details of the study.
- Obtain an informed consent signed and personally dated by the subject or the subject's legally acceptable representative and by the person who conducted the informed consent discussion.
- Obtain the IRB/IEC's written approval/favorable opinion of the written ICF and any other information to be provided to the subjects, prior to the beginning of the study, and after any revisions are completed for new information.

If informed consent is initially given by a subject's legally acceptable representative or legal guardian, and the subject subsequently becomes capable of making and communicating his or her informed consent during the study, consent must additionally be obtained from the subject.

Revise the informed consent whenever important new information becomes available that is relevant to the subject's consent. The investigator, or a person designated by the investigator, should fully inform the subject or the subject's legally acceptable representative or legal guardian, of all pertinent aspects of the study and of any new information relevant to the subject's willingness to continue participation in the study. This communication should be documented.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules applicable to regulatory requirements, the subjects' signed ICF and, in the US, the subjects' signed HIPAA Authorization.

The consent form must also include a statement that BMS and regulatory authorities have direct access to subject records.

For minors, according to local legislation, one or both parents or a legally acceptable representative must be informed of the study procedures and must sign the informed consent form approved for the study prior to clinical study participation. The explicit wish of a minor, who is capable of forming an opinion and assessing this information to refuse participation in, or to be withdrawn from, the clinical study at any time should be considered by the investigator.

Minors who are judged to be of an age of reason must also give their written assent.

Subjects unable to give their written consent (eg, stroke or subjects with or severe dementia) may only be enrolled in the study with the consent of a legally acceptable representative. The subject must also be informed about the nature of the study to the extent compatible with his or her understanding, and should this subject become capable, he or she should personally sign and date the consent form as soon as possible. The explicit wish of a subject who is unable to give his or her written consent, but who is capable of forming an opinion and assessing information to refuse participation in, or to be withdrawn from, the clinical study at any time should be considered by the investigator.

The rights, safety, and well-being of the study subjects are the most important considerations and should prevail over interests of science and society.

### SOURCE DOCUMENTS

The Investigator is responsible for ensuring that the source data are accurate, legible, contemporaneous, original and attributable, whether the data are hand-written on paper or entered electronically. If source data are created (first entered), modified, maintained, archived, retrieved, or transmitted electronically via computerized systems (and/or any other kind of electronic devices) as part of regulated clinical trial activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records (EMRs/EHRs), AE tracking/reporting, protocol required assessments, and/or drug accountability records).

When paper records from such systems are used in place of electronic format to perform regulated activities, such paper records should be certified copies. A certified copy consists of a copy of original information that has been verified, as indicated by a dated signature, as an exact copy having all of the same attributes and information as the original.

#### STUDY TREATMENT RECORDS

Records for study treatments (whether supplied by BMS, its vendors, or the site) must substantiate study treatment integrity and traceability from receipt, preparation, administration, and through destruction or return. Records must be made available for review at the request of BMS/designee or a Health Authority.

| If | Then |
|---|---|
| Supplied by BMS (or its vendors): Records or logs must comply with appli regulations and guidelines and should in | |
| | amount received and placed in storage area |
| | amount currently in storage area |
| | • label identification number or batch number |
| | amount dispensed to and returned by each<br>subject, including unique subject<br>identifiers |
| | amount transferred to another area/site for dispensing or storage |
| | • nonstudy disposition (eg, lost, wasted) |
| | • amount destroyed at study site, if applicable |
| | amount returned to BMS |
| | • retain samples for bioavailability/bioequivalence, if applicable |
| | dates and initials of person responsible for<br>Investigational Product |

| If | Then |
|---|---|
| | dispensing/accountability, as per the Delegation of Authority Form. |
| Sourced by site, and not supplied by BMS or its vendors (examples include IP sourced from the sites stock or commercial supply, or a specialty pharmacy) | The investigator or designee accepts responsibility for documenting traceability and study treatment integrity in accordance with requirements applicable under law and the SOPs/standards of the sourcing pharmacy. These records should include: • label identification number or batch number • amount dispensed to and returned by each subject, including unique subject identifiers • dates and initials of person responsible for Investigational Product dispensing/accountability, as per the Delegation of Authority Form. |

BMS or designee will provide forms to facilitate inventory control if the investigational site does not have an established system that meets these requirements.

### **CASE REPORT FORMS**

An investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation on each individual treated or entered as a control in the investigation. Data that are derived from source documents and reported on the CRF must be consistent with the source documents or the discrepancies must be explained. Additional clinical information may be collected and analyzed in an effort to enhance understanding of product safety. CRFs may be requested for AEs and/or laboratory abnormalities that are reported or identified during the course of the study.

For sites using the Sponsor or designee electronic data capture tool, electronic CRFs will be prepared for all data collection fields except for fields specific to SAEs and pregnancy, which will be reported on the electronic SAE form and paper Pregnancy Surveillance form, respectively. If electronic SAE form is not available, a paper SAE form can be used.

The confidentiality of records that could identify subjects must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

The investigator will maintain a signature sheet to document signatures and initials of all persons authorized to make entries and/or corrections on CRFs.

The completed CRF, SAE/pregnancy CRFs, must be promptly reviewed, signed, and dated by the investigator or qualified physician who is a subinvestigator and who is delegated this task on the Delegation of Authority Form. For electronic CRFs, review and approval/signature is completed electronically through the electronic data capture tool. The investigator must retain a copy of the CRFs including records of the changes and corrections.

Each individual electronically signing electronic CRFs must meet Sponsor or designee training requirements and must only access the electronic data capture tool using the unique user account provided by Sponsor or designee. User accounts are not to be shared or reassigned to other individuals

#### MONITORING

Sponsor or designee representatives will review data centrally to identify potential issues to determine a schedule of on-site visits for targeted review of study records.

Representatives of BMS must be allowed to visit all study site locations periodically to assess the data quality and study integrity. On site they will review study records and directly compare them with source documents, discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable. Certain CRF pages and/or electronic files may serve as the source documents:

In addition, the study may be evaluated by Sponsor or designee internal auditors and government inspectors who must be allowed access to CRFs, source documents, other study files, and study facilities. BMS audit reports will be kept confidential.

The investigator must notify BMS promptly of any inspections scheduled by regulatory authorities, and promptly forward copies of inspection reports to Sponsor or designee.

### RECORDS RETENTION

The investigator must retain all study records and source documents for the maximum period required by applicable regulations and guidelines, or institution procedures, or for the period specified by BMS or designee, whichever is longer. The investigator must contact BMS prior to destroying any records associated with the study.

BMS or designee will notify the investigator when the study records are no longer needed.

If the investigator withdraws from the study (eg, relocation, retirement), the records shall be transferred to a mutually agreed upon designee (eg, another investigator, study site, IRB). Notice of such transfer will be given in writing to BMS or designee.

#### **RETURN OF STUDY TREATMENT**

For this study, study treatments (those supplied by BMS, a vendor or sourced by the investigator) such as partially used study treatment containers, vials and syringes may be destroyed on site.

| If | Then |
|---|---|
| Study treatments supplied by BMS (including its vendors | Any unused study treatments supplied by BMS can only be destroyed after being inspected and reconciled by the responsible Study Monitor unless study treatments containers must be immediately destroyed as required for safety, or to meet local regulations (eg, cytotoxics or biologics). |

| | If study treatments will be returned, the return will be arranged by the responsible Study Monitor. |
|---|---|
| Study treatments sourced by site, not supplied<br>by BMS (or its vendors) (examples include<br>study treatments sourced from the sites stock<br>or commercial supply, or a specialty<br>pharmacy) | It is the investigator's or designee's responsibility to dispose of all containers according to the institutional guidelines and procedures. |

It is the investigator's or designee's responsibility to arrange for disposal, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept. The following minimal standards must be met:

- On-site disposal practices must not expose humans to risks from the drug.
- On-site disposal practices and procedures are in agreement with applicable laws and regulations, including any special requirements for controlled or hazardous substances.
- Written procedures for on-site disposal are available and followed. The procedures must be filed with the site's SOPs and a copy provided to BMS upon request.
- Records are maintained that allow for traceability of each container, including the date disposed of, quantity disposed, and identification of the person disposing the containers. The method of disposal, ie, incinerator, licensed sanitary landfill, or licensed waste disposal vendor must be documented.
- Accountability and disposal records are complete, up-to-date, and available for the Monitor to review throughout the clinical trial period.

It is the investigator's or designee's responsibility to arrange for disposal of all empty containers.

If conditions for destruction cannot be met the responsible Study Monitor will make arrangements for return of study treatments provided by BMS (or its vendors). Destruction of non-study treatments sourced by the site, not supplied by BMS, is solely the responsibility of the investigator or designee.

#### CLINICAL STUDY REPORT AND PUBLICATIONS

A Signatory Investigator must be selected to sign the clinical study report.

For this protocol, the Signatory Investigator will be selected as appropriate based on the following criteria:

- External Principal Investigator designated at protocol development
- National Coordinating Investigator
- Study Steering Committee chair or their designee
- Subject recruitment (eg, among the top quartile of enrollers)
- Involvement in trial design

• Regional representation (eg, among top quartile of enrollers from a specified region or country)

• Other criteria (as determined by the study team)

The data collected during this study are confidential and proprietary to Sponsor or designee. Any publications or abstracts arising from this study must adhere to the publication requirements set forth in the clinical trial agreement (CTA) governing study site or investigator participation in the study. These requirements include, but are not limited to, submitting proposed publications to Sponsor or designee at the earliest practicable time prior to submission or presentation and otherwise within the time period set forth in the CTA.


#### **APPENDIX 3**

ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, FOLLOW-UP, AND REPORTING

#### **ADVERSE EVENTS**

#### **Adverse Event Definition:**

An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered study drug and that does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.

# **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or
  results from other safety assessments (eg, ECG, radiological scans, vital signs
  measurements), including those that worsen from baseline, considered clinically significant
  in the medical and scientific judgment of the investigator Note that abnormal lab tests or
  other safety assessments should only be reported as AEs if the final diagnosis is not
  available. Once the final diagnosis is known, the reported term should be updated to be the
  diagnosis.
- Exacerbation of a chronic or intermittent preexisting condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose, as a verbatim term (as reported by the investigator), should not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae and should specify "intentional overdose" as the verbatim term.

# **Events NOT Meeting the AE Definition**

- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).

### **DEFINITION OF SAE**

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met.

#### SERIOUS ADVERSE EVENTS

# Serious Adverse Event Definition: Any untoward medical occurrence that, at any dose:

Results in death

Is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)

Requires inpatient hospitalization or causes prolongation of existing hospitalization (see note below)

Note: The following hospitalizations are not considered SAEs in BMS clinical studies:

- a visit to the emergency room or other hospital department < 24 hours, that does not result in admission (unless considered an important medical or life-threatening event)
- elective surgery, planned prior to signing consent
- admissions as per protocol for a planned medical/surgical procedure
- routine health assessment requiring admission for baseline/trending of health status (eg, routine colonoscopy)
- medical/surgical admission other than to remedy ill health and planned prior to entry into the study. Appropriate documentation is required in these cases.
- admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (eg, lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason)
- admission for administration of anticancer therapy in the absence of any other SAEs (applies to oncology protocols)

Results in persistent or significant disability or permanent damage

Is a congenital anomaly/birth defect

Is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the subject or may require intervention [eg, medical, surgical] to prevent one of the other serious outcomes listed in the definition above). Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization. Potential drug induced liver injury (DILI) is also considered an important medical event (see Section 8.2.8 for the definition of potential DILI).

Pregnancy and potential DILI must follow the same transmission timing and processes to BMS as used for SAEs (see Section 8.2.6 for reporting pregnancies).

#### **EVALUATING AES AND SAES**

# **Assessment of Intensity**

The intensity of AEs is determined by a physician and will use the following levels:

• Mild: An event that is easily tolerated by the subject, causing minimal discomfort, and not interfering with everyday activities.

- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an even; and both AEs and SAEs can be assessed as severe.

# **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE. A "reasonable possibility of a relationship" conveys that there are facts, evidences, and/or arguments to suggest a causal relationship rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the Investigator's Brochure (IB) and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to Sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to Sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send a SAE follow-up report with the updated causality assessment.

The causality assessment is one of the criteria used when determining regulatory reporting requirements..

# Follow-up of AEs and SAEs

If only limited information is initially available, follow-up reports are required. Note: Follow-up SAE reports must include the same investigator term(s) initially reported.

If an ongoing SAE changes in its intensity or relationship to study drug or if new information becomes available, the SAE report must be updated and submitted within 24 hours to BMS (or designee) using the same procedure used for transmitting the initial SAE report.

All SAEs must be followed to resolution or stabilization.

### REPORTING OF SAES TO SPONSOR OR DESIGNEE

SAEs, whether related or not related to study drug, and pregnancies must be reported to Drug Safety within 24 hours of awareness of the event. SAEs must be recorded on the SAE Report Form. For studies capturing SAEs through electronic data capture (EDC), electronic submission is the required method for reporting. In the event the electronic system is unavailable for transmission, paper forms must be used and submitted immediately. When paper forms are used, the original paper forms are to remain on site. Pregnancies must be recorded on a paper Pregnancy Surveillance Form and transmitted via email or confirmed facsimile (fax) transmission to: **SAE Email Address: SAE Fax Number: Americas: Europe/East Asia Pacific: SAE Telephone Contact** - For questions on SAE/pregnancy reporting, please call: **Americas: Europe/East Asia Pacific:** 


# APPENDIX 4 WOMEN OF CHILDBEARING POTENTIAL DEFINTIONS AND METHODS OF CONTRACEPTION

#### **DEFINITIONS**

### Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

## Women in the following categories are not considered WOCBP

- Premenarchal
- Premenopausal female with 1 of the following:
- Documented hysterectomy
- Documented bilateral salpingectomy
- Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of the subject's medical records, medical examination, or medical history interview.

- Postmenopausal female
  - A postmenopausal state is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.

Note: Females treated with hormone replacement therapy, (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and the investigators should use their judgement in checking serum FSH levels.

• 1 week minimum for vaginal hormonal products (rings, creams, gels)

Approved v3.0

- 4 week minimum for transdermal products
- 8 week minimum for oral products

Other parenteral products may require washout periods as long as 6 months. If the serum FSH level is > 40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal.


# CONTRACEPTION GUIDANCE FOR FEMALE SUBJECTS OF CHILD BEARING POTENTIAL

One of the highly effective methods of contraception listed below is required during study duration and until the end of relevant systemic exposure, defined as 3 days after the end of study treatment, plus 30 days

Local laws and regulations may require use of alternative and/or additional contraception methods.

# **Highly Effective Contraceptive Methods That Are User Dependent**

Failure rate of <1% per year when used consistently and correctly.<sup>a</sup>

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>b</sup>
  - o oral
  - o intravaginal
  - o transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation<sup>b</sup>
  - o oral
  - o injectable

# **Highly Effective Methods That Are User Independent**

- Implantable progestogen-only hormonal contraception associated with inhibition of ovulation<sup>b</sup>
- Intrauterine device (IUD)<sup>c</sup>
- Intrauterine hormone-releasing system (IUS)<sup>c</sup>
- Bilateral tubal occlusion
- Vasectomized partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the subject.

- It is not necessary to use any other method of contraception when complete abstinence is elected.
- WOCBP subjects who choose complete abstinence must continue to have pregnancy tests, as specified in Section 5.1
- Acceptable alternate methods of highly effective contraception must be discussed in the event that the WOCBP subjects chooses to forego complete abstinence

#### **NOTES:**

- Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical studies.
- Hormonal contraception may be susceptible to interaction with the study treatment, which may reduce the efficacy of the contraceptive method. Hormonal contraception is permissible only when there is sufficient evidence that the IMP and other study medications will not alter hormonal exposures such that contraception would be ineffective or result in increased exposures that could be potentially hazardous. In this case, alternative methods of contraception should be utilized.
- Intrauterine devices and intrauterine hormone releasing systems are acceptable methods of contraception in the absence of definitive drug interaction studies when hormone exposures from intrauterine devices do not alter contraception effectiveness

# Less Than Highly Effective Contraceptive Methods That Are User Dependent

Failure rate of > 1% per year when used consistently and correctly.

- Male or female condom with or without spermicide. Male and female condoms cannot be used simultaneously
- Diaphragm with spermicide
- Cervical cap with spermicide
- Vaginal Sponge with spermicide
- Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mechanism of action

### **Unacceptable Methods of Contraception**

- Periodic abstinence (calendar, symptothermal, post-ovulation methods)
- Withdrawal(coitus interruptus).

- Spermicide only
- Lactation amenorrhea method (LAM)

# CONTRACEPTION GUIDANCE FOR MALE SUBJECTS WITH PARTNER(S) OF CHILD BEARING POTENTIAL.

Male subjects with female partners of childbearing potential are eligible to participate if they agree to the following during the treatment and until the end of relevant systemic exposure.

- Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.
- Male subjects are required to use a condom for study duration and until the end of relevant systemic exposure defined as 3 days after the end of treatment in the male subject.
- Female partners of males participating in the study to consider use of effective methods of contraception until the end of relevant systemic exposure, defined as 3 days after the end of treatment in the male subject.
- Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse or use a male condom during each episode of penile penetration during the treatment and until 3 days after the end of treatment.
- Refrain from donating sperm for the duration of the study treatment and for 3 days after the end of treatment.

#### **COLLECTION OF PREGNANCY INFORMATION**

Guidance for collection of Pregnancy Information and outcome of pregnancy on the Pregnancy Surveillance Form is provided in Section 8.2.6 and APPENDIX 3

# APPENDIX 5 STATIC PHYSICIAN'S GLOBAL ASSESSMENT OF PSORIASIS (sPGA)

The static PGA is used to determine the subject's psoriasis lesions overall at a given time point. Overall lesions will be graded for erythema, induration, and scaling based on the scales below. The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score.

| Characteristics | Score | Rating Score |
|---|---|---|
| Erythema (E) (averaged over the whole body) | | <ul> <li>0 = No evidence of erythema, but post inflammatory hyper/hypopigmentation changes may be present</li> <li>1 = Faint erythema</li> <li>2 = Light red coloration</li> <li>3 = Moderate red coloration</li> <li>4 = Bright red</li> </ul> |
| Induration (I) (averaged over the whole body) | | <ul> <li>0 = No evidence of plaque elevation</li> <li>1 = Minimal plaque elevation, barely palpable, = 0.25 mm</li> <li>2 = Mild plaque elevation, slight but definite elevation, indistinct edge, = 0.5 mm</li> <li>3 = Moderate plaque elevation, elevated with distinct edges, = 0.75 mm</li> <li>4 = Severe plaque elevation, hard/sharp borders, ≥ 1 mm</li> </ul> |
| Scaling (S) (averaged over the whole body) | | 0 = No evidence of scaling 1 = Minimal; occasional fine scaling 2 = Mild; fine scale dominates 3 = Moderate; coarse scale predominates 4 = Severe; thick scale predominates |

E + I + S = /3 = (Total Average)

Physician's Static Global Assessment based upon above Total Average

- 0 = Clear, except for residual discoloration
- 1 = Almost clear -majority of lesions have individual scores for E + I + S / 3 that averages 1
- 2 = Mild -majority of lesions have individual scores for E + I + S / 3 that averages 2
- 3 = Moderate majority of lesions have individual scores for E + I + S / 3 that averages 3
- 4 = Severe -majority of lesions have individual scores for E + I + S / 3 that averages 4

Note: Scores should be rounded to the nearest whole number. If total  $\leq 1.49$ , score = 1; if total  $\geq 1.50$ , score = 2.

Clinical Protocol BMS-986165

# APPENDIX 6 PSORIASIS AREA AND SEVERITY INDEX (PASI)

Psoriasis Area and Severity Index (PASI); a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance. Please complete **all** sections of the table and shade in the affected areas on the body diagrams below.

| Dia Oh ava eta vietia | Body region (and weighting factor) | | | | |
|---|---|---|---|---|---|
| Plaque Characteristic Rating score | | Head | Upper Extremities | Trunk | Lower Extremities |
| Erythema (Redness) | 0 = None<br>1 = Slight | | | | |
| Infiltration (Thickness) | 2 = Moderate | | | | |
| Desquamation (Scaling) | 3 = Severe<br>4 = Very severe | | | | |
| Add together each of the | 3 scores for each | of the body regions | to give 4 separate si | ub totals. | • |
| | Sub Totals | A1 = | A2 = | A3 = | A4 = |
| Multiply each sub total by upper extremities, A3 x 0 | | | | | |
| | | A1 x 0.1 = B1 | A2 x 0.2 = B2 | A3 x 0.3 = B3 | A4 x 0.4 = B4 |
| | | B1 = | B2 = | B3 = | B4 = |
| Degree of involvement as % for each body region affected; (score each region with score between 0-6) | 0 = None<br>1 = 1-9 %<br>2 = 10-29%<br>3 = 30-49%<br>4 = 50 -69%<br>5 = 70-89%<br>6 = 90-100% | | | | |
| For each body region multiply sub total B1, B2, B3 and B4 by the <u>score</u> (0-6) of the % of body region involved to give 4 subtotals C1, C2, C3 and C4 | | | | | |
| | | B1 x score = C1 | B2 x score = C2 | B3 x score = C3 | B4 x score = C4 |
| | | C1 = | C2 = | C3 = | C4 = |
| The patient's PASI sco | re is the sum of ( | C1 + C2 + C3 + C4 | | PASI= | |


# APPENDIX 7 SCALP-SPECIFIC PHYSICIAN'S GLOBAL ASSESSMENT (SSPGA)

Please rate overall scalp psoriasis severity by selecting the overall score based on the following rating scale:

| Score | Category | Description |
|---|---|---|
| 0 | Absence of | No evidence of redness, no evidence of thickness, and no |
| | Disease | evidence of scaliness on the scalp |
| | ., | The overall clinical picture consists of flat lesions with barely |
| 1 | Very Mild Disease | perceptible erythema, with or without a trace of overlying fine |
| | | scale |
| 2 | Mild Disease | The overall clinical picture consists of lesions with mild |
| | Willa Discase | erythema, slight, but definite, thickness, and a thin scale layer |
| 3 | Moderate Disease | The overall clinical picture consists of lesions with moderate |
| | Moderate Disease | erythema, a moderate thickness, and a moderate scaled layer |
| | | The overall clinical picture consists of lesions with bright |
| 4 | Severe Disease | erythema, severe thickness, and a severe, coarse thick scale |
| | | layer |





# APPENDIX 9 PHYSICIAN'S GLOBAL ASSESSMENT-FINGERNAILS (PGA-F)

For this assessment in subjects with psoriasis fingernail involvement, the overall condition of the fingernails is rated by the investigator on a 0-4 (5-point) scale. The overall score assigned based on the higher of the nail bed/nail matrix score:

| | | Nail Bed Signs | Nail Matrix Signs |
|---|---|---|---|
| Clear | 0 | Onycholysis- consistent with a normal nail AND Hyperkeratosis- none AND Splinter Hemorrhages-consistent with non-psoriatic splinter hemorrhages | No nonpsoriatic nail plate irregularities including pitting, crumbling, Beau's lines, senile onychorrhexis, and nonpsoriatic leukonychia |
| | | AND Nail Bed Erythema- none | |
| Minimal | 1 | Onycholysis- < 10% involved on all nails OR Hyperkeratosis- present, but barely detectable elevation of nail plate OR Nail Bed Erythema- faint AND Splinter Hemorrhages- consistent with non-psoriatic splinter hemorrhages | No more than 5 pits or psoriatic leukonychia on any nail <b>AND</b> No crumbling |
| Mild | 2 | Onycholysis->10% on five or more nails OR Hyperkeratosis- present with mild elevation of nail plate OR Splinter Hemorrhages- present on four or fewer nails OR Nail Bed Erythema- mild | Five or more nails with mild pitting (eg, >10 pits/nail) or psoriatic leukonychia <b>AND</b> No crumbling |
| Moderate | 3 | Onycholysis->30% on at least one nail OR Hyperkeratosis- present with moderate elevation of nail plate OR Splinter Hemorrhages- scattered and present on five or more nails OR Nail Bed Erythema- moderate | Five or more nails with moderate pitting (eg, >25 pits/nail) AND ≤25% crumbling on any nails |
| Severe | 4 | Onycholysis->50% on at least one nail OR Hyperkeratosis- present with severe elevation of nail plate OR Splinter Hemorrhages- numerous and present on five or more nails OR Nail Bed Erythema- severe | Five or more nails with severe pitting (>50 pits/nail) OR >25% crumbling on any nail |





# APPENDIX 11 PALMOPLANTAR PSORIASIS PHYSICIAN'S GLOBAL ASSESSMENT (pp-PGA)

Palmoplantar (including finger and toe surfaces) psoriasis lesions are evaluated by the investigator based on overall severity, then scored on the following 5-point scale:

| Score | Category | Description |
|---|---|---|
| 0 | Clear | No signs of plaque psoriasis |
| 1 | Almost | Just perceptible erythema and just perceptible scaling |
| | Clear | |
| 2 | Mild | Light pink erythema, with minimal scaling with or without pustules |
| 3 | Moderate | Dull red, clearly distinguishable erythema with diffuse scaling, some thickening of the skin, with or without fissures, with or without pustule formation |
| 4 | Severe | Deep, dark red erythema with obvious and diffuse scaling and thickening as well as numerous fissures with or without pustule formation |




# APPENDIX 13 PSORIASIS SYMPTOMS AND SIGNS DIARY (PSSD)

Please answer each question to the best of your ability. There are no right or wrong answers. Please pay close attention to the time period of interest. These questions ask you to think about the past 24 hours. Please complete the diary at the same time every day.

Individuals with psoriasis may experience a range of symptoms. Please indicate how severe each of the following skin symptoms was in the **past 24 hours**. Please select only one number for each item on the 0 to 10 scale (0=Absent and 10= Worst imaginable).

| Rate the severity of <u>itch</u> in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 2. Rate the severity of dryness in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 3. Rate the severity of <u>cracking</u> in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 4. Rate the severity of skin tightness in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 5. Rate the severity of scaling (build-up of skin) in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 6. Rate the severity of shedding or flaking in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 7. Rate the severity of <u>redness</u> in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 8. Rate the severity of <u>bleeding</u> in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 9. Rate the severity of <u>burning</u> in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst |
| 10. Rate the severity of stinging in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |
| 11. Rate the severity of pain from your psoriasis lesions in the past 24 hours. | 0<br>Absent | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>imaginable |

# APPENDIX 14 DERMATOLOGY LIFE QUALITY INDEX (DLQI)

| Hospital No: | | Date: | | | |
|---|---|---|---|---|---|
| | S | core: | | | |
| Na | ame: D | iagnosis: | | | |
| Αc | ddress: | | | | |
| | ne aim of this questionnaire is to measure to e OVER THE LAST WEEK. Please tick of | • | - | n ha | ns affected your |
| 1. | Over the last week, how itchy, sore, painful or stin been? | <b>ging</b> has your skin | Very<br>much A<br>lot<br>A little | | |
| 2. | Over the last week, how <b>embarrassed</b> or <b>self-cons</b> been because of your skin? | cious have you | Very<br>much A<br>lot<br>A little | | |
| 3. | Over the last week, how much has your skin interfer going <b>shopping</b> or looking after your <b>home</b> or <b>gard</b> | | Very<br>much A<br>lot<br>A little | | Not relevant |
| 4. | Over the last week, how much has your skin influence wear? | ced the <b>clothes</b> you | Very<br>much A<br>lot<br>A little | | Not relevant |
| 5. | Over the last week, how much has your skin affecte leisure activities? | d any <b>social</b> or | Very<br>much A<br>lot<br>A little | | Not relevant |
| 6. | Over the last week, how much has your skin made i any <b>sport</b> ? | t difficult for you to do | Very<br>much A<br>lot<br>A little | | Not relevant |
| 7. | Over the last week, has your skin prevented you from studying? | m <b>working</b> or | y<br>e<br>s | | Not relevant |
| | If "No", over the last week how much has your skin bwork or studying? | oeen a problem at | A<br>lot<br>A<br>littl | | |
| 8. | Over the last week, how much has your skin created your <b>partner</b> or any of your <b>close friends</b> or <b>relativ</b> | | Very<br>much A<br>lot<br>A little | | Not relevant |
| 9. | Over the last week, how much has your skin caused difficulties? | l any <b>sexual</b> | Very<br>much A<br>lot<br>A little | | Not relevant |

Revised Protocol No.: 05 Date: 11-Nov-2020 

| | nical Protocol<br>IS-986165 | IM011065<br>TYK2 Inhibitor | |
|---|---|---|---|
| 10. | Over the last week, how much of a problem has the <b>treatment</b> for your skin been, for example by making your home messy, or by taking up time? | Very<br>much A<br>lot<br>A little | Not relevant |

Please check you have answered EVERY question. Thank you

Revised Protocol No.: 05 Date: 11-Nov-2020


Clinical Protocol IM011065 BMS-986165 TYK2 Inhibitor
























# APPENDIX 20 PSORIATIC ARTHRITIS SCREENING AND EVALUATION (PASE) QUESTIONNAIRE

# PSORIATIC ARTHRITIS SCREENING AND EVALUATION (PASE) QUESTIONNAIRE

Please circle or mark <u>ONLY ONE</u> of the five choices on the following 15 questions. The answers to these questions will help us better understand your symptoms. This should take about 5-6 minutes to complete. Thank you for your time.

| Symptoms sub-scale | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|
| I feel tired for most of the day | 1 | 2 | 3 | 4 | 5 |
| 2. My joints hurt | 1 | 2 | 3 | 4 | 5 |
| 3. My back hurts | 1 | 2 | 3 | 4 | 5 |
| 4. My joints become swollen | 1 | 2 | 3 | 4 | 5 |
| 5. My joints feel 'hot' | 1 | 2 | 3 | 4 | 5 |
| 6. Occasionally, an entire finger or toe becomes swollen, making it look like a 'sausage' | 1 | 2 | 3 | 4 | 5 |
| 7. I have noticed that the pain in my joints moves from one joint to another, eg my wrist will hurt for a few days then my knee will hurt and so on. | 1 | 2 | 3 | 4 | 5 |
| SYMPTOM SCORE (Max 35) | Add scores for questions 1-7 and write in box A | | | | Α. |
| Function sub-scale | Strongly<br>Disagree | Disagree | Neutral | Agree | Strongly<br>Agree |
| 8. I feel that my joint problems have affected my ability to work | 1 | 2 | 3 | 4 | 5 |
| 9. My joint problems have affected my ability to care for myself, eg getting dressed or brushing my teeth | 1 | 2 | 3 | 4 | 5 |
| 10. I have had trouble wearing rings on my fingers or my watch | 1 | 2 | 3 | 4 | 5 |
| 11. I have had trouble getting into or out of a car | 1 | 2 | 3 | 4 | 5 |
| 12. I am unable to be as active as I used to be | 1 | 2 | 3 | 4 | 5 |
| 13. I feel stiff for more than 2 hours after waking up in the morning | 1 | 2 | 3 | 4 | 5 |
| 14. The morning is the worst time of day for me | 1 | 2 | 3 | 4 | 5 |
| 15. It takes me a few minutes to get moving to the best of my ability, any time of the day | 1 | 2 | 3 | 4 | 5 |
| FUNCTION SCORE (Max 40) | Add score box B | B. | | | |


120

| TOTAL PASE SCORE (Max 75) Add scores in boxes A and B and write in box C | C. |
|---|---|
|---|---|

# APPENDIX 21 EIGHT-ITEM PATIENT HEALTH QUESTIONNAIRE (PHQ-8)

The eight-item Patient Health Questionnaire depression scale is established as a valid self-administered diagnostic and severity measure for depressive disorders. It consists of 8 different questions, with an answer scale from 0-3. The overall score is determined by adding up each of the individual answers from each question.

Scoring interpretation is as follows: 0-4 no significant depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately severe depressive symptoms, and 20-24 severe depressive symptoms

# Over the last 2 weeks, how often have you been bothered by any of the following problems?

| | Not at all | Several<br>Days | More than half the days | Nearly<br>every day |
|---|---|---|---|---|
| Little interest or pleasure in doing things | 0 | 1 | 2 | 3 |
| 2. Feeling down, depressed, or hopeless | 0 | 1 | 2 | 3 |
| Trouble falling or staying asleep, or sleeping too much | 0 | 1 | 2 | 3 |
| 4. Feeling tired or having little energy | 0 | 1 | 2 | 3 |
| 5. Poor appetite or over eating | 0 | 1 | 2 | 3 |
| 6. Feeling bad about yourself, or that you are a failure, or have let yourself or your family down | 0 | 1 | 2 | 3 |
| 7. Trouble concentrating on things, such as reading the newspaper, or watching television | 0 | 1 | 2 | 3 |
| 8. Moving or speaking so slowly that other people could have noticed? Or the opposite, being so fidgety or restless that you have been moving around a lot more than usual | 0 | 1 | 2 | 3 |

Total Score:

Clinical Protocol IM011065 BMS-986165 TYK2 Inhibitor

# APPENDIX 22 SUICIDAL IDEATION AND BEHAVIOR CATEGORIES AND DEFINITIONS

#### **Suicidal Ideation**

#### Passive suicidal ideation: wish to be dead

Patient has thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up.

#### Active suicidal ideation: nonspecific (no method, intent, or plan)

General nonspecific thoughts of wanting to end one's life or commit suicide (eg, "I've thought about killing myself") without general thoughts of ways to kill oneself/associated methods, intent, or plan during the assessment period.

# Active suicidal ideation: method, but no intent or plan

Patient has thoughts of suicide and has thought of at least one method during the assessment period. This situation is different than a specific plan with time, place, or method details worked out (eg, thought of method to kill self but not a specific plan). Includes person who would say, "I thought about taking an overdose but I never made a specific plan as to when, where, or how I would actually do it . . . and I would never go through with it."

#### Active suicidal ideation: method and intent, but no plan

Active suicidal thoughts of killing oneself, and patient reports having some intent to act on such thoughts, as opposed to "I have the thoughts but I definitely will not do anything about them."

### Active suicidal ideation: method, intent, and plan

Thoughts of killing oneself with details of plan fully or partially worked out and patient has some intent to carry it out (ie, some degree of intent is implicit in the concept of plan).

#### **Suicidal Behavior**

#### **Completed suicide**

A self-injurious behavior that resulted in fatality and was associated with at least some intent to die as a result of the act. Evidence that the individual intended to kill him- or herself, at least to some degree, can be explicit or inferred from the behavior or circumstance.

#### Suicide attempt

A potentially self-injurious behavior, associated with at least some intent to die as a result of the act. Evidence that the individual intended to kill him- or herself, at least to some degree, can be explicit or inferred from the behavior or circumstance. A suicide attempt may or may not result in actual injury.

# **Interrupted suicide attempt**


Clinical Protocol IM011065 BMS-986165 TYK2 Inhibitor

When the person is interrupted (by an outside circumstance) from starting a potentially self-injurious act (if not for that, actual attempt would have occurred).

# Aborted suicide attempt

When person begins to take steps toward making a suicide attempt, but stops before actually engaging in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops before being stopped by something else.

# Preparatory acts toward imminent suicidal behaviors

This category can include anything beyond a verbalization or thought, but it stops short of a suicide attempt, an interrupted suicide attempt, or an aborted suicide attempt. This might include behaviors related to assembling a specific method (eg, buying pills, purchasing a gun) or preparing for one's death by suicide (eg, giving things away, writing a suicide note).

# **Self-Injurious Behavior Without Suicidal Intent**

Self-injurious behavior associated with no intent to die. The behavior is intended purely for other reasons, either to **relieve** distress (often referred to as self-mutilation (eg, superficial cuts or scratches, hitting or banging, or burns) or to effect change in others or the environment.
